# A Randomized, Controlled, Double-blind, Continuation Study Comparing the Long-term Safety and Efficacy of Orelvo (voclosporin) (23.7 mg Twice Daily) with Placebo in Subjects with Lupus Nephritis

Clinical Protocol Number: AUR-VCS-2016-02

Study Name: AURORA (AURinia Orelvo Renal

Assessments) 2: Aurinia Renal Response in

Lupus with Orelvo (voclosporin)

Date: 21 December 2018

Version Number: 3.0

Previous Protocol Versions: Original V1.0: 13 October 2017

Amendment 1, V2.0: 10 October 2018

IND Number: 114577

EudraCT Number: 2016-004046-28

# NAMES AND ADDRESSES

| | TANIES AND A | IDDRESSES |
|---|---|---|
| Lead Investigator | Name:<br>Address: | |
| | Tel:<br>Fax:<br>Email: | |
| Sponsor | Name:<br>Address: | Aurinia Pharmaceuticals, Inc.<br>#1203 - 4464 Markham Street<br>Victoria, BC<br>V8Z 7X8<br>Canada |
| | Tel:<br>24 Hour: | |
| Clinical Representative | Name:<br>Company:<br>Address: | Aurinia Pharmaceuticals, Inc.<br>#1203 - 4464 Markham Street<br>Victoria, BC<br>V8Z 7X8<br>Canada |
| | Email: | |
| Chief Medical Officer | Name:<br>Company:<br>Address: | Aurinia Pharmaceuticals, Inc.<br>#1203 - 4464 Markham Street<br>Victoria, BC<br>V8Z 7X8<br>Canada |

Email:

Regulatory Representative Name:

Company: Aurinia Pharmaceuticals, Inc. Address: #1203 - 4464 Markham Street

Victoria, BC V8Z 7X8 Canada

Email:

Trial Statistician Name:

Company: Aurinia Pharmaceuticals, Inc. Address: #1203 - 4464 Markham Street

Victoria, BC V8Z 7X8 Canada

Email:

## **DECLARATION OF SPONSOR**

Title: A Randomized, Controlled, Double-blind Continuation Study Comparing the Long-term Safety and Efficacy of Orelvo (voclosporin) (23.7 mg Twice Daily) with Placebo in Subjects with Lupus Nephritis

Version Number/Date: Version 3.0/21 December 2018

This study protocol was subjected to critical review. The information it contains is consistent with current knowledge of the risks and benefits of the study treatment, as well as with the moral, ethical and scientific principles governing clinical research as set out in the Declaration of Helsinki, and the International Council for Harmonisation Guidelines on Good Clinical Practice.

#### Sponsor Representatives

| | () ? DAN 2019 |
|---|---|
| Chief Medical Officer | Date (e.g., DD Month Year) |
| | Date (e.g., DD Month Year) |
| Vice President, Quality and Regulatory<br>Affairs | Date (c.g., DD Month 1 cal) |

# **INVESTIGATOR AGREEMENT FORM**

I have read the attached protocol titled: A Randomized, Controlled, Double-blind Continuation Study Comparing the Long-term Safety and Efficacy of Orelvo (voclosporin) (23.7 mg Twice Daily) with Placebo in Subjects with Lupus Nephritis.

Version Number/Date: Version 3.0/21 December 2018

I agree to comply with the current International Council for Harmonisation Guidelines on Good Clinical Practice and applicable regulations and guidelines.

I agree to ensure that financial disclosure statements will be completed by:

- me (including, if applicable, my spouse (or legal partner) and dependent children);
- my sub-investigators

before the start of the study and to report any changes that affect my financial disclosure status for up to 1 year after the study is completed.

I agree to ensure that the confidential information contained in this document will not be used for any purpose other than the evaluation or conduct of the clinical investigation without the prior written consent of Aurinia Pharmaceuticals Inc.

Signature by the Investigator on this form documents review, agreement and approval of the requirements contained within this protocol.

| Name | |
|-----------|----------------------------|
| Signature | Date (e.g., DD Month Year) |

# **SYNOPSIS**

| Title: | A Randomized, Controlled, Double-blind Continuation Study Comparing the Long-term Safety and Efficacy of Orelvo (voclosporin) (23.7 mg Twice Daily) with Placebo in Subjects with Lupus Nephritis. |
|---|---|
| Short Title: | AURORA (AURinia Orelvo Renal Assessments) 2: Aurinia Renal Response in Lupus Nephritis with Orelvo |
| Study Product: | Orelvo (voclosporin) |
| Indication: | Lupus nephritis |
| Phase: | 3 |
| Sponsor: | Aurinia Pharmaceuticals Inc. |
| Study Code: | AUR-VCS-2016-02 |
| Objectives: | Primary Objective: |
| | • To assess the long-term safety and tolerability of Orelvo compared with placebo for up to an additional 24 months following completion of treatment in the AURORA 1 study in subjects with lupus nephritis (LN). |
| | Secondary Objective: |
| | • To assess the long-term efficacy of Orelvo compared with placebo for up to an additional 24 months following completion of treatment in the AURORA 1 study in subjects with LN. |
| Design: | Prospective, placebo-controlled, double-blind, parallel-group, 24-month continuation study to the AURORA 1 study (AUR-VCS-2016-01). |
| Treatment: | Investigational Treatment: |
| | Orelvo softgel capsules containing 7.9 mg drug. |
| | Subjects who have completed 52 weeks of treatment with study drug and participation in the AURORA 1 study will continue to receive the same treatment as assigned by randomization in the AURORA 1 52-week study (either Orelvo or matching placebo). |
| | Subjects will continue to receive treatment with study drug at the same dose administered at Week 52 of the AURORA 1 study. |
| | After 12 months treatment in the AURORA 2 Continuation Study (i.e., 24 months treatment in total), subjects with controlled UPCR (in the Investigator's opinion), subjects taking the 23.7 mg (3 capsules) twice daily (BID) dose will be permitted to reduce the dose of Orelvo to 15.8 mg (2 capsules) BID if considered appropriate by the Investigator and after consultation with the Medical Monitor. |

Where a dose reduction is considered, the following guidance should be considered:

| AURORA 2: Week 52 Dose | AURORA 2: Reduced Dose |
|---------------------------------|------------------------|
| 23.7 mg BID and UPCR ≥1.5 mg/mg | No reduction |
| 23.7 mg BID and UPCR <1.5 mg/mg | 15.8 mg BID |
| <23.7 mg BID | No reduction |

Notes: BID = Twice daily; UPCR = Urine protein creatinine ratio

For any subject receiving an Orelvo (or matching placebo) dose of <23.7 mg BID and presenting with 2 consecutive clinically relevant (in the opinion of the investigator) increases in urine protein creatinine ratio (UPCR), a dose increase of voclosporin (to a maximum of 23.7 mg BID) or appropriate rescue therapy per the Investigator's discretion and current treatment guidelines should be considered.

All subjects will continue to receive background therapy of mycophenolate mofetil (MMF) and oral corticosteroids, if applicable, starting at the same dose as at the end of the AURORA 1 study. When clinically indicated, subjects are allowed to be completely titrated off of oral corticosteroids; the sites will contact the Medical Monitor if the dose of oral corticosteroids is to be increased.

#### Inclusion Criteria:

- 1. Written informed consent before any study-specific procedures are performed.
- 2. Male or female subjects who have completed 52 weeks of treatment with study drug in the AURORA 1 study. Subjects who had a temporary interruption and successfully restarted study drug during the AURORA 1 study will be allowed with Medical Monitor approval.
- 3. In the opinion of the Investigator, subject requires continued immunosuppressive therapy.
- 4. Women of childbearing potential must continue to use effective contraception and have a negative urine pregnancy test at Month 12. Two effective forms of contraception must be used simultaneously unless abstinence is the chosen method. Subjects must use effective contraception during the study (see Section 5.4, Adequate/Effective Contraception).
- 5. Subject is willing to continue taking oral MMF for the duration of the study.

#### **Exclusion Criteria:**

- 1. Subjects unable or unwilling to give written informed consent and/or to comply with study procedures.
- 2. Currently taking or known need for any of the medications or food items listed in Section 7.8, Prohibited Therapy and Concomitant Treatment during the study.
- 3. Subjects currently requiring renal dialysis (hemodialysis or peritoneal dialysis) or expected to require dialysis during the study period.
- 4. A planned kidney transplant within study treatment period.
- Subjects with any medical condition which, in the Investigator's judgment, may be associated with increased risk to the subject or may interfere with study assessments or outcomes.

| | 6. Subjects who are pregnant, breast feeding or, if of childbearing potential, not using adequate contraceptive precautions. |
|---|---|
| | 7. Vaccines using live organisms, virus or bacterial, while taking the study treatment. |
| Primary Endpoint: | Adverse events (AE) profile and routine biochemical and hematological assessments. |
| Secondary | Proportion of subjects in renal response defined as: |
| Endpoints: | <ul><li>UPCR of ≤0.5 mg/mg</li></ul> |
| | <ul> <li>estimated glomerular filtration rate (eGFR) ≥60 mL/min/1.73 m<sup>2</sup></li> <li>or no confirmed decrease from baseline in eGFR of &gt;20%</li> </ul> |
| | <ul> <li>Received no rescue medication for LN</li> </ul> |
| | <ul> <li>Did not receive more than 10 mg prednisone for ≥3 consecutive<br/>days or for ≥7 days in total during the 8 weeks prior to the renal<br/>response assessment.</li> </ul> |
| | • Subjects who withdraw from the study prior to the response assessment will be defined as non-responders. |
| | • Proportion of subjects in partial renal response defined as a 50% reduction from baseline in UPCR. |
| | Renal flare as adjudicated by the Clinical Endpoints Committee (CEC). |
| | Extra-renal flare as adjudicated by the CEC. |
| | SELENA-SLEDAI scores by visit. |
| | • Change in UPCR, eGFR, urine protein, and serum creatinine from AURORA 1 baseline. |
| | • Change in immunology parameters (complement 3 (C3), complement 4 (C4), and antidoublestranded deoxyribonucleic acid (DNA)) from AURORA 1 baseline. |
| | • Change in health-related quality of life (HRQoL) (SF-36) from AURORA 1 baseline. |
| | Healthcare Resource Utilization (HRU). |

#### Procedures: See Schedule of Events for full details of protocol required procedures and applicable visits (and timings). Subjects who have completed 52 weeks of treatment with study drug in the AURORA 1 study and have provided signed and dated informed consent will be entered into this study. Subjects meeting the required eligibility criteria will be registered in the interactive web response system for the AURORA 2 continuation study, using the same subject number assigned in the AURORA 1 study. Subjects will continue to receive either Orelvo or matching placebo as randomized in the AURORA 1 study. Study drug treatment in the continuation study will remain blinded. Dosing of Orelvo or matching placebo in AURORA 2 is detailed in the Treatment section above. All subjects will continue to receive background therapy of MMF andoral corticosteroids, if applicable, starting at the same dose as at the end of the AURORA 1 study. When clinically indicated, subjects are allowed to be completely titrated off of oral corticosteroids; the sites will contact the Medical Monitor if the dose of oral corticosteroids is to be increased. All subjects will receive up to 24 additional months of treatment, i.e., maximum 36 months in total (12 months in AURORA 1 plus 24 months in AURORA 2). After 12 months treatment in the AURORA 2 Continuation Study (i.e., 24 months treatment in total), subjects with controlled UPCR (in the Investigator's opinion), taking the 23.7 mg (3 capsules) BID dose will be permitted to reduce the dose of Orelvo to 15.8 mg (2 capsules) BID if considered appropriate and at the discretion of the Investigator and after consultation with the Medical Monitor. Subjects who permanently discontinue treatment with study drug will be treated at the Investigator's discretion, and where appropriate in accordance with current guidelines (e.g., American College of Rheumatology (ACR 2012)). Subjects will return for all remaining study visits and assessments unless they have withdrawn consent. Those subjects who have withdrawn consent to complete remaining visits will be advised to return for the End of Treatment/Early Termination Visit. All subjects will have a safety follow-up visit after the last dose of study drug, and an assessment of vital status at 6 and 12 months post study. Sample Size: Subjects will enter this protocol from the AURORA 1 study in order to provide the opportunity of an additional 24 months of treatment (total

36 months of treatment); no sample size calculation is required.

Statistical Methods:

Analysis:

All statistical summaries and analyses will be undertaken at study closure once the last subject has completed the Visit 24 safety follow-up visit. A complete description of the statistical analyses to be performed will be presented in a Statistical Analysis Plan (SAP).

The study will incorporate an unblinded, interim analysis of both safety and efficacy data. The timing of this interim analysis is expected to be 3 months post the final subject final visit of the AURORA 1 study (i.e., when the last subject reaches Visit 16 of the AURORA 2 continuation study).

#### Populations:

The safety analysis set will consist of all subjects who receive at least 1 dose of study drug in the continuation study.

The efficacy analysis set will be based on the intent-to-treat (ITT) principles and will consist of all consented subjects.

#### Safety Endpoints:

The analysis and summary of the safety endpoints will be conducted on the safety set.

Adverse events will be aggregated by System Organ Class and preferred term and presented as summary tables.

Laboratory values (based on results from the central laboratory), vital signs and other safety parameters will be summarized by visit as absolute values and change from AURORA 1 baseline. Laboratory values outside of defined normal ranges will be summarized.

#### **Efficacy Endpoints:**

All the secondary efficacy analyses will be performed on the ITT set. Data for each visit (as well as change from AURORA 1 study baseline as required) will be summarized by treatment group and visit for each secondary endpoint.

The following key secondary efficacy endpoints will be analyzed using the ITT population using logistic regression with terms for treatment group, baseline UPCR, biopsy class and MMF use at baseline (from AURORA 1) in the model.

- Proportion of subjects in renal response at Months 12, 18, 24, 30, and 36.
- Proportion of subjects in partial renal response at Months 12, 18, 24, 30, and 36.

The results will be expressed as an odds ratio (and associated two sided 95% confidence interval [CI]) for Orelvo compared to placebo. Odds ratios greater than unity show the odds of response are greater for Orelvo than for placebo and therefore indicate a benefit of the Orelvo treatment arm.

The proportion of subjects with renal and extra-renal flares (as adjudicated by the CEC) will be analyzed in a similar fashion to the proportion of subjects achieving response.

The following secondary endpoints will be analyzed using a Mixed Effect Model Repeated Measures (MMRM). The MMRM model will include terms for treatment, visit, treatment by visit interaction, and baseline. Results will be expressed as differences between treatment arms (along with the associated 95% CI).

- Change in UPCR, eGFR, urine protein, and serum creatinine from AURORA 1 baseline at each visit.
- Change in immunology parameters (C3, C4, and anti-dsDNA) from AURORA 1 baseline at each visit.

- Change in HRQoL (SF-36) from AURORA 1 baseline at Months 12, 18, 24, 30, and 36.
- Change in SELENA-SLEDAI scores by visit at Months 12, 18, 24, and 36.

Healthcare Resource Utilization at Months 12, 15, 18, 21, 24, 27, 30, 33, and 36. Key aspects will be summarized by visit and changes over time will be explored.

# **SCHEMA**



Notes: BID = Twice daily; IV = Intravenous; MMF = Mycophenolate mofetil.

# **AUR-VCS-2016-02 SCHEDULE OF EVENTS**

| Visit (1) | Visit 15<br>(End of<br>Treatment<br>Visit of<br>AURORA<br>1) <sup>(1)</sup> (2) | Visit 16 | Visit 17 | Visit 18 | Visit 19 | Visit 20 | Visit 21 | Visit 22 | Visit 23 End of Study/ Early Terminatio n(3) | Visit 24<br>Safety<br>Follow-up <sup>(4)</sup> |
|---|---|---|---|---|---|---|---|---|---|---|
| Month <sup>(5)</sup> | 12<br>±10 days | 15<br>±10 days | 18<br>±10 days | 21<br>±10 days | 24<br>±10 days | 27<br>±10 days | 30<br>±10 days | 33<br>±10 days | 36<br>±10 days | 37<br>±10 days |
| Informed consent | <b>√</b> | | | | | | | | | |
| Eligibility criteria | ✓ | | | | | | | | | |
| Physical examination <sup>(6)</sup> | ( <b>√</b> ) | | | | | | | | <b>√</b> | |
| Vital signs<br>(BP, pulse,<br>temperature) | (4) | <b>√</b> | <b>√</b> | <b>√</b> | <b>√</b> | <b>~</b> | <b>√</b> | <b>✓</b> | <b>√</b> | <b>√</b> |
| Kidney<br>Biopsy <sup>(7)</sup> | | , | / | | | | | | | |
| ECG <sup>(8)</sup> | (✓) | | ✓ | | ✓ | | | | ✓ | |
| Laboratory<br>assessments <sup>(</sup> | (✓) | <b>√</b> | <b>~</b> | <b>~</b> | <b>√</b> | <b>~</b> | <b>~</b> | <b>√</b> | <b>√</b> | <b>✓</b> |
| Serum<br>pregnancy<br>test <sup>(10)</sup> | ( <b>∀</b> ) | | | | <b>√</b> | | | | ✓ | |

| Visit (1) | Visit 15<br>(End of<br>Treatment<br>Visit of<br>AURORA<br>1) <sup>(1) (2)</sup> | Visit 16 | Visit 17 | Visit 18 | Visit 19 | Visit 20 | Visit 21 | Visit 22 | Visit 23 End of Study/ Early Terminatio n(3) | Visit 24<br>Safety<br>Follow-up <sup>(4)</sup> |
|---|---|---|---|---|---|---|---|---|---|---|
| Month <sup>(5)</sup> | 12<br>±10 days | 15<br>±10 days | 18<br>±10 days | 21<br>±10 days | 24<br>±10 days | 27<br>±10 days | 30<br>±10 days | 33<br>±10 days | 36<br>±10 days | 37<br>±10 days |
| Urine pregnancy test <sup>(11)</sup> | <b>√</b> | <b>√</b> | <b>✓</b> | <b>✓</b> | | <b>~</b> | <b>~</b> | <b>√</b> | | |
| AEs <sup>(12)</sup> | (✓) | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ |
| Concomitant medications <sup>(</sup> | (✓) | <b>√</b> | <b>✓</b> | ✓ | <b>~</b> | <b>~</b> | <b>√</b> | ✓ | ✓ | <b>√</b> |
| Study<br>treatment<br>dispensing<br>and<br>compliance | <b>√</b> | <b>√</b> | <b>√</b> | <b>~</b> | ~ | <b>~</b> | <b>~</b> | <b>~</b> | <b>√</b> (14) | |
| MMF<br>dispensing | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | <b>√</b> | ✓ | |
| Oral<br>corticosteroi<br>ds <sup>(15)</sup> | <b>√</b> | ✓ | ✓ | <b>√</b> | <b>~</b> | ✓ | <b>√</b> | ✓ | | |
| Urinalysis | (✓) | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ |
| FMV urine collection | (✓) | <b>√</b> | <b>√</b> | <b>√</b> | <b>√</b> | <b>√</b> | <b>√</b> | <b>√</b> | <b>√</b> | <b>√</b> |

| Visit (1) | Visit 15<br>(End of<br>Treatment<br>Visit of<br>AURORA<br>1) <sup>(1)</sup> (2) | Visit 16 | Visit 17 | Visit 18 | Visit 19 | Visit 20 | Visit 21 | Visit 22 | Visit 23 End of Study/ Early Terminatio n(3) | Visit 24 Safety Follow-up <sup>(4)</sup> |
|---|---|---|---|---|---|---|---|---|---|---|
| Month <sup>(5)</sup> | 12<br>±10 days | 15<br>±10 days | 18<br>±10 days | 21<br>±10 days | 24<br>±10 days | 27<br>±10 days | 30<br>±10 days | 33<br>±10 days | 36<br>±10 days | 37<br>±10 days |
| 24-hour urine (16) | (✔) | | <b>√</b> | | <b>√</b> | | ✓ | | <b>√</b> | |
| SELENA-<br>SLEDAI | (✓) | | ✓ | | ✓ | | | | ✓ | |
| Health–<br>related QoL<br>(SF-36) <sup>(17)</sup> | (✓) | | <b>~</b> | | <b>√</b> | | <b>√</b> | | <b>√</b> | |
| HRU <sup>(18)</sup> | (✓) | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | ✓ | |

- 1 Month 12 Visit refers to the End of Treatment Visit 15 of the AURORA 1 (AUR-VCS-2016-01) study.
- 2 Visit 15 assessments marked (-) will be provided from the results of the Week 52 Visit in the AURORA study.
- 3 Subjects who discontinue therapy will attend their regularly scheduled study visits to the end of the study. Subjects who withdraw consent and terminate the study early should be advised to attend both Visit 23 and the Safety Follow-up Visit (Visit 24).
- 4 Subjects will have a safety follow-up visit after the last dose of study drug, and an assessment of vital status at 6 and 12 months post study.
- 5 Unscheduled visits/assessments can be done as needed. AEs, concomitant medications and verbal compliance check should be completed.
- 6 Abbreviated physical examination only required. Height is not required.
- 7 At sites that are able to meet the biopsy requirements,
- 8 During the study, in the event that a subject is noted to have a QTcF value exceeding 500 msec, or >60 msec more than baseline, the ECG will be repeated; see Section 9.1.4.1, Procedures to Manage a Treatment-Emergent Increase in QTc.
- 9 Laboratory assessments will be performed according to the schedule in Section 9.1.1, Laboratory Assessments; subjects will be fasting for 8 hours on the day of study entry on Month 12 (Week 52/ End of Treatment Visit of the AURORA 1 study) and at Month 24 and Month 36 End of Study visit.
- 10 Serum pregnancy test to be evaluated at central laboratory at Month 12 using AURORA 1 Visit 15 result, Month 24, and Month 36.
- 11 Urine pregnancy test to be performed at Month 12 (AURORA 1 Visit 15) for subjects who consent for enrollment into the AURORA 2 continuation study. In addition, urine pregnancy tests to be performed at all other visits indicated (except Month 24 and Month 36 where serum pregnancy test is performed).
- 12 AEs will be recorded after the subject signs the ICF.
- 13 Concomitant medications include all herbal medicines and supplements taken by the subject.
- 14 Compliance only.
- 15 All subjects will continue to receive oral corticosteroids starting at the same dose as at the end of the AURORA 1 study. When clinically indicated, subjects are allowed to be completely titrated off of oral corticosteroids; the sites will contact the Medical Monitor if the dose of oral corticosteroids is to be increased.
- 16 24-hour urine collection should begin 2 days prior to the scheduled study visit in order not to coincide with the FMV sampling due on the day of the study visit.
- 17 For details on HRQoL assessments (SF-36), see Section 9.3.1, Health-related Quality of Life Assessments (HRQoL).
- 18 For details on Healthcare Resource Utilization, see Section 9.3.2, Healthcare Resource Utilization Assessment.

Abbreviations: AE=adverse event; BP=blood pressure; ECG=electrocardiogram; FMV=first morning void; HRU = healthcare resource utilization; ICF=informed consent form; LN=lupus nephritis; MMF=mycophenolate mofetil; QTcF=QT interval duration corrected for heart rate using method of Fridericia; SAE=serious adverse event; SELENA-SLEDAI=Safety of Estrogens in Lupus Erythematosus National Assessment - Systemic Lupus Erythematosus Disease Activity Index; SLE=systemic lupus erythematosus.

# TABLE OF CONTENTS

| | Page |
|---|---|
| NAMES AND ADDRESSES | 2 |
| DECLARATION OF SPONSOR | 4 |
| INVESTIGATOR AGREEMENT FORM | 5 |
| SYNOPSIS | |
| SCHEMA | |
| AUR-VCS-2016-02 SCHEDULE OF EVENTS | |
| TABLE OF CONTENTS | 17 |
| LIST OF TABLES | 22 |
| LIST OF APPENDICES | 22 |
| LIST OF ABBREVIATIONS | 23 |
| 1. INTRODUCTION AND BACKGROUND | 26 |
| 1.1 Background of the Disease and Treatment Options – Lupus Nephritis | |
| 1.1.1 Limitations of Current Treatment | |
| 1.2 Rationale for the Use of Calcineurin Inhibitors in Lupus Nephritis | 28 |
| 1.2.1 Mechanism of Action | 28 |
| 1.2.2 Use of Immunosuppression in Lupus Nephritis | 28 |
| 1.2.3 Clinical Studies of Calcineurin Inhibitors in Lupus Nephritis | 29 |
| 1.2.4 Voclosporin | |
| 1.2.4.1 Pharmacokinetic Considerations | |
| 1.2.4.2 Lupus Nephritis Clinical Development | |
| 1.2.5 Potential Toxicities | 32 |
| 2. RATIONALE | 34 |
| 2.1 Dose Rationale | 34 |
| 3. STUDY OBJECTIVES | 36 |
| 3.1 Primary Objective | |
| 3.2 Secondary Objective | |
| 3.3 Endpoints | |
| 3.3.1 Primary Endpoint | |
| 3.3.2 Secondary Endpoints | |
| 3.3.2.1 Key Secondary Endpoints | 36 |
| 3.3.2.2 Other Secondary Endpoints | |
| 3.3.2.3 | 37 |

| 4. | INVESTIGATIONAL PLAN | 38 |
|---|---|---|
| 4.1 | Overall Study Design | 38 |
| 4.2 | Duration of Subject Participation and Study | 38 |
| 5. | SELECTION, WITHDRAWAL OF SUBJECTS AND PERMANE | ENT |
| | DISCONTINUATION OF DRUG | 39 |
| 5.1 | Number of Subjects | 39 |
| 5.2 | Inclusion Criteria | 39 |
| 5.3 | Exclusion Criteria | 39 |
| 5.4 | Adequate/Effective Contraception | 40 |
| 5.5 | Withdrawal of Subjects | 40 |
| 5.6 | Discontinuation of Study Treatment | 41 |
| 5.6. | Discontinuation from Study Treatment Due to Renal Flare or Non-response to | |
| | Therapy | |
| 5.6.2 | Discontinuation of Study Treatment Due to an Adverse Event | 41 |
| 6. | RANDOMIZATION, BLINDING AND UNBLINDING PROCEDURES | 42 |
| 6.1 | Randomization | |
| 6.2 | Blinding | 42 |
| 6.3 | Unblinding | |
| 7. | STUDY TREATMENTS | 43 |
| 7.1 | Dosage Forms/Formulation | |
| 7.1. | | |
| 7.1.2 | · | |
| 7.1.3 | Background Therapy | 43 |
| 7.1.3 | | |
| 7.1.3 | | |
| 7.2 | Drug Dosage and Administration | 43 |
| 7.2. | Treatment Arms | 43 |
| 7.2.2 | 2 Dosing Guidelines | 44 |
| 7.2.2 | 2.1 Orelvo/Placebo – Study Treatment | 44 |
| 7.2.2 | 2.2 Corticosteroids | 45 |
| 7.2.2 | 2.3 Mycophenolate Mofetil (Background Therapy) | 45 |
| 7.3 | Package and Labeling | 46 |
| 7.4 | Study Treatment Allocation | 46 |
| 7.5 | Site Supply, Storage, Accountability | 46 |
| 7.5. | Site Supply | 46 |
| 7.5.2 | 2 Storage | 46 |
| 7.5.3 | 3 Accountability | 47 |
| 7.6 | Orelvo/Placebo Dose Modification | |
| 7.6. | Deterioration in Renal Function | 48 |

| 7.6.1.1 Decrease in eGFR >30% and eGFR <60 mL/min/1.73 m <sup>2</sup> | 48 |
|-----------------------------------------------------------------------|----|
| 7.6.1.2 Decrease in eGFR ≤30% and eGFR <60 mL/min/1.73 m <sup>2</sup> | 48 |
| 7.6.1.3 Decrease in eGFR ≤20% | 49 |
| 7.6.1.4 Decrease in eGFR >30% and eGFR ≤90 mL/min/1.73 m <sup>2</sup> | 49 |
| 7.6.1.5 Decrease in eGFR >30% and eGFR >90 mL/min/1.73 m <sup>2</sup> | 49 |
| 7.6.1.6 Recovery of eGFR | 49 |
| 7.7 Procedures for Overdose | 49 |
| 7.8 Prohibited Therapy and Concomitant Treatment | 49 |
| 7.8.1 Prohibited Medications | |
| 7.8.2 Allowed Concomitant Medications | 51 |
| 7.9 Increased Blood Pressure | 51 |
| 8. RISKS/PRECAUTIONS | 52 |
| 9. STUDY PROCEDURES | 53 |
| 9.1 Description of Study Assessments | 53 |
| 9.1.1 Laboratory Assessments | 53 |
| 9.1.1.1 | 55 |
| 9.1.2 Physical Examinations | 55 |
| 9.1.3 Vital Signs | 56 |
| 9.1.3.1 Blood Pressure Management | 56 |
| 9.1.4 Standard 12-lead Electrocardiogram | 56 |
| 9.1.4.1 Procedures to Manage a Treatment-Emergent Increase in QTc | 57 |
| 9.1.5 Lupus Disease Activity Assessments | 57 |
| 9.1.6 Kidney Biopsy | 57 |
| 9.2 Schedule of Assessments | 57 |
| 9.2.1 Screening Visit Procedures | 58 |
| 9.2.2 Treatment Procedures | 58 |
| 9.2.3 End of Study (or Early Discontinuation) Procedures | 60 |
| 9.2.4 Follow-up Procedures | 60 |
| 9.2.5 Unscheduled Visit | 61 |
| 9.3 Study Specific Assessment Procedures | 62 |
| 9.3.1 Health-related Quality of Life Assessments (HRQoL) | 62 |
| 9.3.1.1 Short Form Health Survey (SF-36) | 62 |
| 9.3.2 Healthcare Resource Utilization (HRU) Assessment | 62 |
| 10. EVALUATION, RECORDING AND REPORTING OF AES AND SAES | |
| 10.1 Definitions | |
| 10.1.1 Adverse Event | |
| 10.1.2 Adverse Drug Reaction | |
| 10.1.3 Serious Adverse Event | |
| 10.1.4 Suspected Unexpected Serious Adverse Reaction | 64 |

| 10.2 Adverse Event Descriptors | 64 |
|-------------------------------------------------------|----|
| 10.2.1 Intensity/Severity Categorization | 64 |
| 10.2.2 Causal Relationship Categorization | 65 |
| 10.2.3 Outcome Categorization | 65 |
| 10.2.4 Symptoms of the Disease Under Study | 65 |
| 10.2.5 Clinical Laboratory Evaluations | 66 |
| 10.2.6 Abuse, Misuse, Overdose and Medication Error | 66 |
| 10.3 Reporting Procedure for AEs, SAEs, and Pregnancy | |
| 10.3.1 Adverse Events | 66 |
| 10.3.2 Serious Adverse Events | 67 |
| 10.3.3 Pregnancy | 69 |
| 11. CLINICAL ENDPOINTS COMMITTEE | 70 |
| 12. DATA AND SAFETY MONITORING BOARD PROCED | |
| 13. STATISTICAL ANALYSIS | 72 |
| 13.1 Statistical Methods | 72 |
| 13.2 Sample Size and Power Calculations | 72 |
| 13.3 Populations | 72 |
| 13.3.1 Intent-to-Treat Set | 72 |
| 13.3.2 Safety Set | 72 |
| 13.4 Background and Demographic Characteristics | 72 |
| 13.5 Study Treatment | 72 |
| 13.6 Concomitant Therapy | 73 |
| 13.7 Endpoint Evaluations | 73 |
| 13.7.1 Primary Safety Endpoint | 73 |
| 13.7.2 Secondary Efficacy Endpoints | 73 |
| 13.7.2.1 Key Secondary Efficacy Endpoints | 73 |
| 13.7.2.2 Other Secondary Efficacy Endpoints | |
| 13.7.2.3 | 74 |
| 13.8 Statistical and Analytical Methods | 74 |
| 13.8.1 Safety Analysis | |
| 13.8.2 Efficacy Analysis | |
| 13.8.2.1 Response Endpoints | |
| 13.8.2.2 Renal flare and Extra-renal flare | |
| 13.8.2.3 Change from Baseline Endpoints | |
| 13.8.2.4 Healthcare Resource Utilization (HRU) | |
| 13.9 Safety Evaluations | |
| 13.10 Interim Analyses | |
| 13.11 Other Evaluations | 76 |
| 14. ETHICAL CONDUCT OF THE STUDY | 77 |

| 14.1 Informed Consent | 77 |
|----------------------------------------------|----------------------------|
| 14.2 Institutional Review Board or EC/IEC | 77 |
| 15. QUALITY CONTROL AND QUALITY | ASSURANCE78 |
| 16. ADMINISTRATIVE PROCEDURES | 79 |
| 16.1 Sponsor's Responsibilities | 79 |
| 16.1.1 Study Supplies | 79 |
| 16.1.2 Insurance | 79 |
| 16.1.3 Study Monitoring | 79 |
| 16.2 Investigator's Responsibilities | 80 |
| 16.2.1 Reporting and Recording of Data | 80 |
| 16.2.2 Investigator Training | 80 |
| 16.2.3 Source Documentation | 80 |
| 17. PROCEDURE FOR MODIFICATION | N OF PROTOCOL OR PREMATURE |
| TERMINATION OF THE STUDY | 82 |
| 17.1 Protocol Waivers, Deviations and Violat | ions82 |
| 17.2 Study Termination | 82 |
| 18. POLICY FOR PUBLICATION AND PR | RESENTATION OF DATA83 |
| 19. REFERENCES | 84 |

# LIST OF TABLES

| | Page |
|---|---|
| Table 1 | Review of Laboratory Assessments |
| LIST OF APPENDICES | |
| | Page |
| Appendix 1 | Drug Therapy for the Treatment of Hypertension87 |
| Appendix 2 | Measurement of Blood Pressure |
| Appendix 3 | International Society of Nephrology and the Renal Pathology Society (ISN/RPS) 2003 Classification of Lupus Nephritis89 |
| Appendix 4 | 1997 Update of the 1982 American College of Rheumatology Revised Criteria for the Classification of Systemic Lupus Erythematosus91 |
| Appendix 5 | Systemic Lupus Erythematosus Disease Activity Measure (SELENA-SLEDAI) |
| Appendix 6 | Expanded List of Allowed Concomitant Medications95 |
| Appendix 7 | Summary of Treatment and Food Restrictions |
| Appendix 8 | Short Form Health Survey (SF-36) HRQoL Assessment98 |
| Appendix 9 | 104 |

#### LIST OF ABBREVIATIONS

ACE Angiotensin converting enzyme

ACR American College of Rheumatology

ADR Adverse drug reaction

AE Adverse event

ALMS Aspreva Lupus Management Study

ANC Absolute neutrophil count

ARB Angiotensin II receptor blocker

AUC $_{0-12}$  Area under the curve between 0 and 12 hours

AURA-LV Aurinia Urinary protein Reduction Active – Lupus with

Voclosporin

Aurinia Aurinia Pharmaceuticals Inc.

AURION Aurinia early Urinary protein ReductION Predicts Response

AURORA AURinia Orelvo Renal Assessments

AZA Azathioprine

BID Twice daily

BP Blood pressure

C3 / C4 Complement 3 / complement 4

CEC Clinical Endpoints Committee

CI Confidence interval

CKD-EPI Chronic Kidney Disease Epidemiology Collaboration

C<sub>max</sub> Maximum concentration

CNI Calcineurin inhibitor

CsA Cyclosporine A

CYP3A4/5 Cytochrome P450 3A4/5

DNA deoxyribonucleic acid

dsDNA Double-stranded deoxyribonucleic acid

DSMB Data and Safety Monitoring Board

EC Ethics Committee

EDC Electronic data capture

ECG Electrocardiogram

eCRF Electronic case report form

eGFR Estimated glomerular filtration rate

ESRD End-stage renal disease

FMV first morning void

GCP Good Clinical Practice

GI Gastrointestinal

GMP Good Manufacturing Practice

HCP Health care professional

HR Heart rate

HRQoL Health-related quality of life

HRU Healthcare Resource Utilization

IB Investigator's Brochure

ICF Informed consent form

ICH International Council for Harmonisation

IEC Independent Ethics Committee

IRB Institutional Review Board

IRT Interactive Response Technologies

ITT Intent-to-treat

IV Intravenous

IVC Intravenous cyclophosphamide

LN Lupus nephritis

MMF Mycophenolate mofetil

MMRM Mixed Effect Model Repeated Measures

NSAID Non-steroidal anti-inflammatory drug

Orelvo Voclosporin (for Phase 3 lupus nephritis indication)

P-gp P-glycoprotein

PK Pharmacokinetic

QTc Corrected QT interval

QTcF QT interval duration corrected for heart rate using method of

Fridericia

SAE Serious adverse event

SAP Statistical analysis plan

SELENA Safety of Estrogens in Lupus Erythematosus National Assessment

SF-36 36-Item Short Form Health Survey

SLE Systemic lupus erythematosus

SLEDAI Systemic Lupus Erythematosus Disease Activity Index

 $t_{1/2}$  Terminal elimination half-life

TEAE Treatment-emergent adverse event

UPCR Urine protein creatinine ratio

WHO World Health Organization

## 1. INTRODUCTION AND BACKGROUND

# 1.1 Background of the Disease and Treatment Options – Lupus Nephritis

Lupus nephritis (LN) is the most common serious manifestation of systemic lupus erythematosus (SLE). Lupus nephritis is divided into different classes according to the level of treatment required, using a classification system for renal biopsy pathology originally developed by the World Health Organization (WHO). The classification of LN has evolved and the "International Society of Nephrology/Renal Pathology Society 2003 Classification of Lupus Nephritis" is now widely used and has a higher level of inter-observer reproducibility than the original classification (see Appendix 3). For subjects with Class III, IV (proliferative), or V (membranous), or combinations of these forms of LN, the standard of care is treatment with corticosteroids and immunosuppressive therapy.

Lupus nephritis manifests as diverse patterns of immune complex-mediated renal disease affecting glomerular, tubulointerstitial, and vascular compartments. It can lead to permanent and irreversible tissue damage within the kidney, resulting in end-stage renal disease (ESRD), and thus making LN a serious and potentially life-threatening condition. In subjects with LN, renal damage results in proteinuria and/or hematuria and a decrease in renal function as evidenced by reduced creatinine clearance and estimated glomerular filtration rate (eGFR), and increased serum creatinine levels.

In LN as in other serious renal diseases, the main clinical outcomes are progression to ESRD (i.e., the need for long-term dialysis or transplantation) and death. The current standard of care for LN, corticosteroids and immunosuppressants, has improved the prognosis of the disease considerably. Incidence rates of ESRD in LN, however, appear to have been stable over recent years, possibly reflecting the limits of effectiveness of current treatments or lack of adherence to treatments by subjects. The most recent studies have reported 10-year survival rates of over 90% and, although the overall risk of developing ESRD in subjects with LN is approximately 15%, the 5-year risk of developing ESRD has been found to be as low as 5% [1]. Recently, 10-year follow-up data of LN subjects treated with intravenous cyclophosphamide (IVC) for active disease followed by maintenance treatment with azathioprine (AZA) found rates of ESRD to be approximately 7% [2].

#### 1.1.1 Limitations of Current Treatment

The current treatment paradigm for LN includes 2 goals, based on the severity of disease. The first goal of treatment in subjects with LN is intended to bring the disease under control as quickly as possible to limit the potential for extensive renal scarring or loss of life. This phase of treatment is particularly critical for those subjects at highest risk for ESRD (i.e., subjects with clinical or laboratory indicators of active nephritis, such as biopsy evidence of

proliferative nephritis, active urinary sediment, elevated serum creatinine, and/or proteinuria). In subjects with severe LN, the achievement of complete or partial remission, as demonstrated by stabilization or improvement in renal function, improvement in proteinuria, and normalization of active urinary sediment, has been shown to be associated with better patient and renal survival. Treatment of LN (i.e., induction treatment) typically consists of high doses of both corticosteroids and immunosuppressants.

The second goal of treatment, after the patient successfully responds to treatment, is to maintain remission by preventing renal flares and any resulting deterioration in renal function. In this second phase of treatment, lower doses of both corticosteroids and immunosuppressants are used.

Corticosteroids are the cornerstone of treatment in SLE and have been the standard since the 1950s to treat both renal and non-renal manifestations. Intravenous (IV) steroid pulse therapy is widely used to rapidly treat relapsing LN but does not provide longterm management. Oral corticosteroids taken for prolonged periods and at high doses are often needed, but have potentially severe, and at times irreversible adverse effects including risk of infection, hyperlipidemia, hypertension, osteoporosis, diabetes, and accelerated atherosclerosis. Induction treatment recommendations advocate the use of immunosuppressants in conjunction with high-dose oral corticosteroids, to enable a rapid taper to a lower maintenance dose of steroids. Steroid-sparing therapies are needed in order to- treat disease activity and also minimize cumulative and high-dose steroid exposure.

Intravenous cyclophosphamide, while classically considered the standard of care for induction therapy, is still associated with significant potentially life-threatening toxicities, such as the increased risk of severe infections including sepsis, malignancy, and major morbidity, such as permanent gonadal failure.

Recent studies have shown that induction treatment with mycophenolate mofetil (MMF) has similar efficacy to that of IVC. The authors of a recent meta-analysis concluded that MMF is as efficacious as IVC and is not associated with the risk of infertility, which is a significant toxicity of IVC in this patient population [3]. In the Aspreva Lupus Management Study (ALMS), a comparison of MMF and IVC in the treatment of active LN, 50.4% subjects with active LN entering the study had nephrotic-range proteinuria (>3 g/day) [4]. Intravenous cyclophosphamide and MMF reduced proteinuria to a similar extent. However, even after 24 weeks of therapy with either MMF or IVC in the setting of a clinical study, subjects had substantial residual proteinuria. At the end of 24 weeks of therapy, normal (<500 mg/24 hours) protein excretion levels were observed in only 27% of subjects who received IVC and 23.8% of subjects who received MMF [5]. The findings from ALMS indicate that there exists a substantial unmet medical need for more effective treatments for active LN with heavy proteinuria.

The importance of proteinuria and reduction of proteinuria as prognostic factors for renal flares, ESRD and death in subjects with LN is well documented. Proteinuria in itself is related to progression of renal disease through effects on the glomerulus and tubulointerstitium [6]. In observational studies, proteinuria has been shown to be a predictor of adverse renal outcomes, cardiovascular disease, and mortality in subjects with non-diabetic proteinuric nephropathies [7].

# 1.2 Rationale for the Use of Calcineurin Inhibitors in Lupus Nephritis

#### 1.2.1 Mechanism of Action

Calcineurin inhibitors (CNIs) are a class of immunosuppressants which reversibly inhibit immunocompetent lymphocytes, particularly T-lymphocytes in the  $G_0$  and  $G_1$  phase of the cell-cycle, and also reversibly inhibit the production and release of lymphokines. Voclosporin, a CNI, mediates its suppressive effects by binding to a ubiquitous intracellular protein cyclophilin. This complex, in turn, inhibits the calcium- and calmodulin-dependent serine/threonine phosphatase activity of the enzyme calcineurin. Calcineurin inhibition then prevents the activation of various transcription factors necessary for the induction of cytokine genes during T-cell activation, such as interleukin-2, interleukin-4, tumor necrosis factor- $\alpha$ , granulocytemacrophage- colony stimulating factor, and interferon- $\gamma$ .

## 1.2.2 Use of Immunosuppression in Lupus Nephritis

Calcineurin inhibitors are standard treatment to prevent acute rejection in subjects who have received transplants. Since the development of cyclosporine in the early 1980s, standard immunosuppression regimens to prevent rejection post-transplantation have included steroids and a CNI; more recently other immunosuppressants, such as MMF, have been added to standard therapy. The rationale for use of CNIs in autoimmune diseases include potent effects on T-cell activation and immunomodulatory effects. ATcell mediated immune response is an important feature of the pathogenesis of many of these diseases, including LN. Calcineurin inhibitors also have specific anti-proteinuric effects. The podocyte is a key cell in the glomerular capillary wall that maintains the integrity of the filtration barrier and prevents the development of proteinuria in healthy individuals, while being the primary target of injury in proteinuric- kidney disease. Podocyte injury is an important factor in the progression of LN. It typically occurs due to immune complex deposition but may also occur in the absence of this histologic feature [8]. Podocyte function depends on a complex and unique structure that, in turn, depends on a tightly regulated actin cytoskeleton. Synaptopodin acts as a key stabilizer of the actin cytoskeleton in podocytes. When synaptopodin is phosphorylated, it binds to another protein, 14-3-3, and is thus protected from degradation. Calcineurin dephosphorylates synaptopodin allowing its degradation, thus promoting proteinuria by destabilization of the podocyte actin cytoskeleton. Expression of activated calcineurin in podocytes leads to proteinuria. By inhibiting activated calcineurin, tacrolimus thus exerts a specific

anti-proteinuric effect by preventing the degradation of the podocytestabilizing protein -synaptopodin. Taken together, these data suggest that the anti-proteinuric effects of CNIs may be explained by their direct effect on the podocyte actin cytoskeleton as well as immunomodulatory effects on T-lymphocytes [9].

## 1.2.3 Clinical Studies of Calcineurin Inhibitors in Lupus Nephritis

Bao et al, 2008 [10] performed an open-label study in 40 subjects with Class V+IV LN. Subjects were randomized to either IVC and prednisolone or "multi-target therapy" with MMF plus tacrolimus (4 mg/day) and prednisolone. In the multi-target group, 50% achieved complete remission compared with 5% in the standard IVC group at 6 months. Estimated glomerular filtration rate normalized in both groups, but there was a significantly larger reduction in proteinuria in the multi-target therapy group.

Miyasaka et al, 2009 [11] evaluated the efficacy and safety of tacrolimus in 63 subjects receiving glucocorticoid therapy for LN in a double-blind, placebo-controlled, randomized trial. Subjects with persistent nephritis requiring 10 mg/day prednisone were randomized to receive 28 weeks of treatment with tacrolimus (3 mg/day) or placebo. There was a statistically significant improvement in the primary endpoint, the Lupus Nephritis Disease Activity Index, in the tacrolimus group compared to the placebo group. Daily urinary protein excretion (the percentage of subjects with urine protein <0.3 g/day at the final evaluation) also showed a significant decrease in the tacrolimus group. However, measures of glucose intolerance were more frequent in tacrolimus-treated subjects. The authors concluded that tacrolimus should be considered one of the options to treat LN. On the basis of the results of this study, tacrolimus was approved for the treatment of LN in Japan.

In an observational study conducted by Cortes-Hernandez et al, 2010 [12], 70 subjects who had received MMF as continuous therapy were followed over a 5-year period. Tacrolimus was added as rescue therapy in 17 subjects who were treatment failures or had renal flares on treatment with MMF. The authors reported a significant reduction in proteinuria at 3 months, and after 2 years of follow-up, it was concluded that tacrolimus was a safe and effective treatment for MMF non-responsive cases.

Several smaller pilot studies and case series in subjects with LN, including subjects with membranous nephropathy, have suggested a treatment benefit of tacrolimus with or without MMF [13-19].

The available data suggest a plausible mechanism of action by which CNIs may provide treatment benefits in LN. The clinical evidence is suggestive of improvement in measures of response in active LN and improvement in extrarenal manifestations of SLE and immunologic parameters.

#### 1.2.4 Voclosporin

Voclosporin is a next-generation CNI developed for the treatment of autoimmune diseases and for use in the prevention of organ graft rejection. Voclosporin is structurally similar to cyclosporine A (CsA) except for a novel modification of a functional group on the amino acid 1 residue of the molecule. This alteration has changed the binding of voclosporin to calcineurin leading to a 3- to 5-fold increase in potency when compared to CsA. This modification has also shifted metabolism away from amino acid 1, the major site of metabolism for CsA, thus altering the metabolic profile. This in turn has led to faster elimination of metabolites resulting in lower measured metabolite exposure as compared to CsA. The combination of increased potency and decreased measured metabolite exposure, for voclosporin as compared to CsA, has led to better pharmacokinetic (PK)/ pharmacodynamic predictability.

During the development of this investigational product the legacy names of voclosporin, VCS, are referenced in discussions related to historical usage. However, for the LN Phase 3 clinical development program, the name of the investigational product will be referred to as Orelvo, the proposed trade name. These legacy names should all be considered interchangeable unless specifically identified as different.

Prior to the LN clinical development program, approximately 2,200 subjects received investigational products containing voclosporin in 14 Phase 1 and 10 Phase 2/3 clinical studies in the indications of transplant rejection, psoriasis and non-infectious uveitis. An overview of the data for these clinical studies are presented in the Investigator's Brochure (IB).

#### 1.2.4.1 Pharmacokinetic Considerations

Voclosporin approximates linear multiexponential PKs. Exposure to voclosporin was dose-related with maximum concentrations occurring  $\leq 2$  hours with a terminal elimination half-life ( $t_{1/2}$ ) of  $\geq 30$  hours. Drug accumulation was minor with accumulation factors of approximately 2 hours after twice daily (BID) dosing. Administration of voclosporin oral solution with either low- or high-fat meals decreased both the rate and extent of absorption which appeared to be related to the fat content of the meal. It is therefore recommended that Orelvo (voclosporin) be administered on an empty stomach to ensure adequate absorption.

Voclosporin has been shown to be a substrate of cytochrome P450 3A4/5 (CYP3A4/5). Concomitant administration of ketoconazole, a strong CYP3A4/5 inhibitor, led to a 6-fold increase in maximum concentration (C<sub>max</sub>) and an 18-fold increase in area under the curve between 0 and 12 hours (AUC<sub>0-12</sub>) for voclosporin. Concomitant administration of rifampin, an inducer of CYP3A4/5, resulted in a decrease in exposure to voclosporin. Maximum concentration decreased approximately 70%, the area under the concentration curve decreased approximately 90%, and t<sub>1/2</sub> decreased 85%. Consequently, both ketoconazole and rifampin are contraindicated with Orelvo (voclosporin). Concomitant administration of voclosporin and

midazolam, a model substrate of CYP3A4/5 and potential inhibitor of CYP3A4/5, did not result in statistically significant changes in the rate or extent of exposure to midazolam or  $\alpha$ -hydroxymidazolam-.

Voclosporin is both a substrate for and an inhibitor of P-glycoprotein (P-gp). Concomitant administration of verapamil, a known inhibitor of P-gp, demonstrated an approximate 3-fold increase in C<sub>max</sub> and AUC<sub>0-12</sub> of voclosporin. Concomitant administration of digoxin, a P-gp substrate, resulted in statistically significant increases in digoxin C<sub>max</sub> and area under the curve between 0 and 24 hours (AUC<sub>0-24</sub>) and a decrease in clearance. Therefore, concomitant administration of P-gp substrates with voclosporin would be expected to result in increased exposure to the substrate. Clinicians are advised to consider the benefit/risk of concomitant P-gp substrate drugs carefully.

## 1.2.4.2 Lupus Nephritis Clinical Development

The AURA-LV study (Protocol AUR-VCS-2012-01) was a randomized, controlled, double-blind Phase 2 study comparing the efficacy and safety of voclosporin (23.7 mg BID or 39.5 mg BID) with placebo in achieving remission in patients with active LN. All patients received background therapy with MMF and corticosteroid taper. The duration of the study was 48 weeks with 265 subjects randomized; the study has completed. The primary endpoint of complete remission was defined as: urine protein creatinine ratio (UPCR) of  $\leq$ 0.5 mg/mg at 24 weeks (using first morning void [FMV]) and eGFR  $\geq$ 60 mL/min/1.73 m² or no confirmed decrease from baseline in eGFR of  $\geq$ 20%. In addition, patients could not receive rescue medications for LN (defined as >10 mg prednisone/day for >3 consecutive days or >7 days total from Weeks 16-24) to be considered for complete remission.

The 24-week primary endpoint assessment for the AURA-LV clinical study demonstrated that the groups were generally well balanced for age, gender and race, with a trend to higher proteinuria and lower eGFR data in the low-dose voclosporin arm. The low dose achieved a statistically significant benefit over placebo for the primary efficacy assessment of complete remission at 24 weeks (odds ratio (OR) [95% confidence intervals [CI]] = 2.03, [1.01, 4.05], p=0.045), without a statistically significant improvement seen in the high dose. The results were confirmed by 24-hour urine collections (p=0.047). Both the low- and high-dose voclosporin were statistically superior to placebo in partial remission, time to complete remission, and time to partial remission. A mean reduction in serum creatinine was seen in both arms (0.2 mg/dL low, 0.1 high; p<0.001). In the voclosporin groups, eGFR fell by a median of 8-9 mL/min by Week 4 and then stabilized over the course of the study. Blood pressure (BP) did not vary by group. The correlation of 24-hour urine protein and using the FMV was assessed from the results of the AURA-LV study demonstrating a high degree of correlation (Pearson Correlation Coefficient = 0.92).

Over 90% of subjects experienced at least 1 adverse event (AE); the most common being infectious disease (56.2% low-dose, 63.6% high-dose and 50.0% placebo), GI disorders (41.6% low-dose, 52.3% high-dose and 36.4% placebo). More serious adverse events (SAEs) occurred in the voclosporin groups (25.8% low-dose, 25.0% high-dose, 15.8% placebo), and were consistent with those observed in LN patients. There were 13 (4.9%) deaths during the study. There were more deaths in the voclosporin low-dose arm (10) than in either the voclosporin high-dose (2) or placebo (1) arms, with the majority (11/13) occurring in Asia. All deaths were assessed by the Investigators as unrelated to study treatment.

In summary, no new or unexpected safety signals were observed with the use of voclosporin in LN subjects; voclosporin was generally well tolerated over a 48-week period. The overall safety profile is consistent with the expectations for the class of drug, the patient population, and concomitant therapies.

The AURION study (protocol AUR-VCS-2014-01) was an exploratory open-label Phase 2 study assessing the short-term predictors of remission of voclosporin 23.7 mg BID in combination with standard of care in patients with active LN. All subjects received background therapy with MMF and corticosteroids. The duration of the study was 48 weeks with 10 subjects randomized; the study has completed. The AURION study showed that 7 (70.0%) subjects showed early UPCR reduction of at least 25% from baseline while 4 (40.0%) subjects had early normalization of anti-dsDNA and 2 (20.0%) subjects each showed early normalization of C3 and C4 at Week 8. The results suggest that a combination of early reduction of UPCR and early normalization of complement C3 and C4 may be useful in predicting response. Treatment with voclosporin 23.7 mg BID in combination with MMF and corticosteroids resulted in complete remission in 7/10 (70.0%) subjects at 24 weeks and 4/8 (50.0%) subjects at 48 weeks. Improvements in UPCR, anti-dsDNA, C3, C4, urine protein, and serum albumin levels from baseline were observed during treatment, with stable GFR. These findings suggest that voclosporin in combination with MMF and corticosteroids is beneficial for patients with active LN. No new or unexpected safety signals were observed with the use of voclosporin in LN patients; voclosporin was well-tolerated over a 48-week period. The overall safety profile was consistent with the expectations for the class of drug, the patient population, and concomitant therapies.

#### 1.2.5 Potential Toxicities

Voclosporin has been studied in numerous disease states. When examining LN, there were a small proportion of voclosporin treated subjects that experienced an early drop of  $\geq 30\%$  in eGFR, however that proportion then remains stable over time. None of these treatment-emergent adverse events (TEAEs) were classed as serious. The majority of TEAEs of decreased GFR were classed as mild or moderate, and resulted in permanent discontinuation of study drug in 1 (1.1%) placebo subject, 7 (7.9%) voclosporin low-dose subjects and

5 (5.7%) voclosporin high-dose subjects. There were more TEAEs of hypertension seen in the voclosporin-treated patients compared to placebo however, overall mean systolic and diastolic BP decreased in all groups, without statistically significant differences seen between groups. Overall, only 1 (1.1%) subject, in the voclosporin high-dose group, had a TEAE of hypertension that resulted in permanent discontinuation of study drug.

There was evidence of an increased incidence of TEAEs over placebo and with increased dose of voclosporin in the System Organ Classes of Infections and Infestations, Gastrointestinal (GI) Disorders, and Vascular Disorders.

There were more deaths in the voclosporin low-dose arm (10) than in either the voclosporin high-dose (2) or placebo (1) arms, with the majority (11/13) occurring in South-East Asia. All deaths were assessed by the Investigator and Data and Safety Monitoring Board (DSMB) as unrelated to study treatment. A full description of AEs can be found in the IB.

## 2. RATIONALE

The rationale for the development of Orelvo and the choice of doses is to introduce a novel CNI to the LN patient population, with meaningful efficacy while minimizing toxicities common to other CNIs. In clinical studies, a favorable efficacy/safety profile for Orelvo has been demonstrated in the prevention of renal transplant rejection.

As evaluated in nonclinical and clinical studies (healthy volunteers, moderate to severe psoriasis, renal transplantation, and uveitis) Orelvo is well tolerated and exhibits AEs that are typical of other CNIs yet seen to a lesser extent than that seen historically with other CNIs.

The aim of the Phase 3 continuation study (AURORA 2) is to assess the long-term safety and tolerability of Orelvo, added to the standard of care treatment in LN, for an additional 24 months, following a treatment period of 52 weeks in the AURORA 1 study (AUR-VCS-2016-01). All subjects will continue to receive background therapy of MMF and oral corticosteroids, if applicable, starting at the same dose as at the end of the AURORA 1 study. When clinically indicated, subjects are allowed to be completely titrated off of oral corticosteroids; the sites will contact the Medical Monitor if the dose of oral corticosteroids is to be increased. Subjects with LN, who have completed 52 weeks of treatment with study drug in the AURORA 1 study, will be eligible to enter the study; subjects who had a temporary interruption and successfully restarted study drug during the AURORA 1 study will be allowed with Medical Monitor approval. The long-term safety and tolerability of the drug combination will be assessed from its safety profile while demonstrating the continued ability to achieve and maintain long-term renal response, by reducing the level of proteinuria (as measured by UPCR), for up to an additional 24 months. The primary endpoint of the AURORA 2 study will be the AE profile and biochemical and hematological assessments at 24 months.

#### 2.1 Dose Rationale

The AURORA 2 study is designed to evaluate the safety and tolerability of Orelvo 23.7 mg BID versus placebo, for an additional 24 months following a treatment period of 52 weeks in the AURORA 1 study. Orelvo and/or placebo are herein referred to as study treatment. Subjects will continue to receive the same treatment as assigned by randomization in the AURORA 1 52-week study (either Orelvo or matching placebo). Subjects will continue to receive treatment with study drug at the same dose administered at Week 52 of the AURORA 1 study (see Section 7, Study Treatments).

Orelvo 23.7 mg BID will continue to be administered as a fixed dose without the use of therapeutic drug monitoring. After 12 months treatment in the AURORA 2 Continuation Study (i.e., 24 months treatment in total), subjects with controlled UPCR (in the Investigator's opinion), taking the 23.7 mg (3 capsules) BID dose will be permitted to reduce the dose of

Orelvo to 15.8 mg (2 capsules) BID if considered appropriate and at the discretion of the Investigator and after consultation with the Medical Monitor.

Population PK analyses of voclosporin concentrations from the clinical development program (including healthy subjects, subjects with renal impairment, subjects with hepatic impairment, renal transplant, and plaque psoriasis) demonstrated that weight did not have a significant effect on the PKs of voclosporin. The protocol contains provisions for management of dose based on safety concerns, in particular, BP and renal function. The safety data from the use of voclosporin demonstrates that these risks are dose-related, reversible, and can be managed by dose reduction and temporary interruption.

#### 3. STUDY OBJECTIVES

# 3.1 Primary Objective

• To assess the long-term safety and tolerability of Orelvo compared with placebo for up to an additional 24 months following completion of treatment in the AURORA 1 study in subjects with LN.

# 3.2 Secondary Objective

 To assess the long-term efficacy of Orelvo compared with placebo for up to an additional 24 months following completion of treatment in the AURORA 1 study in subjects with LN.

# 3.3 Endpoints

# 3.3.1 Primary Endpoint

• AE profile and routine biochemical and hematological assessments.

# 3.3.2 Secondary Endpoints

## 3.3.2.1 Key Secondary Endpoints

- Proportion of subjects in renal response defined as:
  - UPCR of  $\leq 0.5$  mg/mg
  - eGFR ≥60 mL/min/1.73 m<sup>2</sup> or no confirmed decrease from baseline in eGFR of >20%
  - Received no rescue medication for LN (see Section 7.8, Prohibited Therapy and Concomitant Treatment)
  - Did not receive more than 10 mg prednisone for ≥3 consecutive days or for
     ≥7 days in total during the 8 weeks prior to the renal response assessment.
- Subjects who withdraw from the study prior to the response assessment will be defined as non-responders.
- Proportion of subjects in partial renal response defined as a 50% reduction from baseline in UPCR.
- Renal flare as adjudicated by the Clinical Endpoints Committee (CEC).
- Extra-renal flare as adjudicated by the CEC.
- SELENA-SLEDAI scores by visit.
- Change in UPCR, eGFR, urine protein, and serum creatinine from AURORA 1 baseline.

## 3.3.2.2 Other Secondary Endpoints

- Change in immunology parameters (C3, C4, and anti-dsDNA) from AURORA 1 baseline.
- Change in health-related quality of life (HRQoL) (SF-36) from AURORA 1 baseline.
- Healthcare Resource Utilization (HRU).



## 4. INVESTIGATIONAL PLAN

## 4.1 Overall Study Design

This is a Phase 3, randomized, prospective, placebo-controlled, double-blind, parallel-group, 24-month continuation study to the AURORA 1 study (AUR-VCS-2016-01). Subjects who have completed 52 weeks of treatment with study drug in the AURORA 1 study and meet all of the inclusion criteria and none of the exclusion criteria will be eligible to consent into the study.

Using an Interactive Response Technologies (IRT) system, eligible subjects will commence dosing with either oral Orelvo or matching placebo, as randomized into AURORA 1, at the same dose as was given at the time of completion of the AURORA 1 study, using the same subject number, for up to 24 additional months, i.e., maximum 36 months in total (12 months in AURORA 1 plus 24 months in AURORA 2). After 12 months treatment in the AURORA 2 Continuation Study (i.e., 24 months treatment in total), subjects with controlled UPCR (in the Investigator's opinion) taking the 23.7 mg BID dose will be permitted to reduce the dose of Orelvo to 15.8 mg BID, if considered appropriate and at the discretion of the Investigator and after consultation with the Medical Monitor. All subjects will continue to receive background therapy of MMF and oral corticosteroids, if applicable, starting at the same dose as at the end of the AURORA 1 study. When clinically indicated, subjects are allowed to be completely titrated off of oral corticosteroids; the sites will contact the Medical Monitor if the dose of oral corticosteroids is to be increased (see Section 7.2.2.2, Corticosteroids and Section 7.2.2.3, Mycophenolate Mofetil (Background Therapy)).

Assessments at Month 12 will be provided from the results of the Week 52/ End of Treatment Visit in the AURORA 1 study (AUR-VCS-2016-01). All subjects will return for assessment of safety and efficacy in Months 15, 18, 21, 24, 27, 30, 33, and 36. See Schedule of Events, for detailed information regarding visits.

All subjects, completed or withdrawn, will complete the End of Treatment/Early Termination assessments (Visit 23) at Month 36 or at the time of early termination. All subjects will have a safety follow-up visit (Visit 24) at Month 37 after the last dose of study drug, to collect any new AEs and concomitant medications. At the follow-up visit, UPCR and eGFR will be assessed as well. An assessment of vital status will occur at 6 and 12 months post study. For subject withdrawal procedures and criteria, see Section 5.5, Withdrawal of Subjects.

# 4.2 Duration of Subject Participation and Study

The expected duration of subject participation is approximately 25 months. An assessment of vital status will occur at 6 and 12 months post study. The treatment duration is 24 months with a further follow-up visit 4 weeks after last dose (completion or early termination).

# 5. SELECTION, WITHDRAWAL OF SUBJECTS AND PERMANENT DISCONTINUATION OF DRUG

## 5.1 Number of Subjects

Subjects will consent to enter this protocol from the AURORA 1 study and will continue to receive treatment with study drug at the same dose administered at Week 52 of the AURORA 1 study.

#### 5.2 Inclusion Criteria

The following inclusion criteria must be met for each subject:

- 1. Written informed consent before any study-specific procedures are performed.
- 2. Male or female subjects who have completed 52 weeks of treatment with study drug in the AURORA 1 study. Subjects who had a temporary interruption and successfully restarted study drug during the AURORA 1 study will be allowed with Medical Monitor approval.
- 3. In the opinion of the Investigator, subject requires continued immunosuppressive therapy.
- 4. Women of childbearing potential must continue to use effective contraception and have a negative urine pregnancy test at Month 12. Two effective forms of contraception must be used simultaneously unless abstinence is the chosen method. Subjects must use effective contraception during the study (see Section 5.4, Adequate/Effective Contraception).
- 5. Subject is willing to continue taking oral MMF for the duration of the study.

#### 5.3 Exclusion Criteria

- 1. Subjects unable or unwilling to give written informed consent and/or to comply with study procedures.
- 2. Currently taking or known need for any of the medications or food items listed in Section 7.8, Prohibited Therapy and Concomitant Treatment during the study.
- 3. Subjects currently requiring renal dialysis (hemodialysis or peritoneal dialysis) or expected to require dialysis during the study period.
- 4. A planned kidney transplant within study treatment period.
- Subjects with any medical condition which, in the Investigator's judgment, may be associated with increased risk to the subject or may interfere with study assessments or outcomes.

- 6. Subjects who are pregnant, breast feeding or, if of childbearing potential, not using adequate contraceptive precautions.
- 7. Vaccines using live organisms, virus or bacterial, while taking the study treatment.

## 5.4 Adequate/Effective Contraception

Women of childbearing potential must have a negative urine pregnancy test at Month 12. Two effective forms of contraception must be used simultaneously unless abstinence is the chosen method. Effective contraception must be used before beginning study treatment, during study dosing, and for 6 weeks following discontinuation of study treatment or MMF dosing, even when there has been a history of infertility, unless due to surgical sterilization. Women not of childbearing potential are defined as women without menses for at least 12 consecutive months or surgically sterilized.

Sexually active men, both reproductively competent and vasectomized, are required to use condoms during treatment and for at least 90 days after cessation of study treatment or MMF. In addition, female partners of male subjects are recommended to use an effective contraception during their partner's treatment and for at least 90 days after the last dose of study treatment or MMF. Male subjects are to refrain from making sperm donations during treatment and for at least 90 days after cessation of study treatment or MMF.

An effective and medically acceptable method of birth control means the chance of pregnancy, when using that type of birth control, is less than 1% per year if used correctly. These birth control methods (i.e., reliable forms of contraception) include birth control pills (combined oral contraceptives), hormone implants, hormone shots, and some intrauterine contraceptive devices. The use of MMF in this study can also reduce the effectiveness of the oral contraceptive pill.

Barrier methods (e.g., condoms, diaphragm, or cervical cap/sponge) when used alone are not considered highly effective.

Although abstinence, when adhered to, is an effective method of birth control, other additional effective contraception methods should be used where there is any doubt. The method of contraception needs to be discussed with the Investigator throughout the study period in order to confirm the method used is considered effective.

# 5.5 Withdrawal of Subjects

Subjects may voluntarily withdraw from study participation at any time for any reason. Alternatively, subjects may be withdrawn at the Investigator's discretion if it is in the subject's best interest.

Every effort should be made for subjects who withdraw from the study, either voluntarily or at the Investigator's discretion, to undergo end of study assessments (Visit 23), if possible. If possible, the subject should also be advised to come for the Safety Follow-up Visit 4 weeks after last dose (Visit 24). If a subject refuses end of study procedures, the reason for refusal should be fully documented in the subject's source document and recorded in the study specific electronic case report form (eCRF). It is the subject's right to withdraw from the study without providing a reason. In this case, the source documents and the eCRF should document the reason for discontinuation as "withdrawal of consent." Withdrawn subjects will not be replaced.

# 5.6 Discontinuation of Study Treatment

Discontinuation of study treatment does not necessarily constitute withdrawal from the study.

If any subject is discontinued from study treatment, the reason for discontinuation will be documented in the eCRF. If the reason for discontinuing study treatment is an AE or an abnormal laboratory test result, the specific event or test will be recorded in the eCRF. Except for cases involving pregnancy, subjects who are discontinued from study treatment should undergo all study visits and assessments up to and including Month 36 or Early Termination Visit – Visit 23, if possible. All subjects that discontinue study treatment should attend at least 1 further assessment after the last dose of study drug. Guidance on when study treatment must be discontinued is in Section 7.6, Orelvo/Placebo Dose Modification.

# 5.6.1 Discontinuation from Study Treatment Due to Renal Flare or Non-response to Therapy

If the subjects require treatment with IV methylprednisolone or any rescue medication other than that permitted in the protocol (see Section 7.2.2.2, Corticosteroids), they should be permanently discontinued from the study treatment and will be considered a treatment failure. Subjects who are permanently discontinued from study treatment will be treated as deemed appropriate by the Investigator.

## 5.6.2 Discontinuation of Study Treatment Due to an Adverse Event

Subjects may be permanently discontinued from study treatment because of the appearance of an unacceptable AE. It is vital to obtain follow-up data on any subject withdrawn because of an AE. In any case, every effort must be made to evaluate protocol-specified safety follow-up procedures (see Section 10.3, Reporting Procedure for AEs, SAEs, and Pregnancy). If a subject is withdrawn due to an AE, the event should be followed by the Investigator through contact with the subject until resolution or stabilization has occurred. All AEs should be followed until resolution, stabilization or the subject is lost to follow-up and cannot be contacted.

## 6. RANDOMIZATION, BLINDING AND UNBLINDING PROCEDURES

## 6.1 Randomization

On the Month 12 visit (Week 52/ End of Treatment Visit of AURORA 1 study), subjects meeting the required eligibility criteria will continue to receive either oral Orelvo 23.7 mg BID or matching placebo, as randomized in the AURORA 1 study. Subjects will be allocated the same subject number assigned in the AURORA 1 study.

All subjects enrolled must be identifiable throughout the study. The Investigator will maintain a list of subject numbers and subject names to enable records to allow subject numbers to be linked to patient medical records, if required.

## 6.2 Blinding

Study drug treatment in the continuation study will remain blinded.

In order to preserve the double-blind design, subjects that consented to the placebo group will be matched to the active dosage groups. Dosing schedule in the placebo group will be the same as that of the active treatment group. To this end, the double-blind nature of this study preserves the blind with respect to active study treatment and placebo.

All study personnel and subjects will be blinded to the study treatment administered during the study. Orelvo and placebo will be identical in taste, smell, and appearance. The site staff, monitors, and study subjects will remain blinded until the end of the study. In case of emergency, the unblinding process below should be followed.

# 6.3 Unblinding

In the rare event that an AE or pregnancy occurs for which knowledge of the identity of the study treatment administered is necessary to manage the subject's condition, the IRT code for that subject may be broken and the test substance identified. Procedures for unblinding will be provided in a separate manual.

Should emergency unblinding be required, the Investigator should call the

Medical Monitor before unblinding wherever possible; however, the
Investigator is responsible for the medical care of the individual study subject, and does not
require the agreement of the Medical Monitor before unblinding. The reason for unblinding
must be documented. The information on study treatment should only be used for decision
making in the subject's further treatment. Details on unblinded treatment assignments should
not be shared with the Study Monitor and project team.

#### 7. STUDY TREATMENTS

## 7.1 Dosage Forms/Formulation

All study treatment to be used in this study will be manufactured in accordance with current Good Manufacturing Practice (GMP). Study treatment will be supplied by Aurinia.

## 7.1.1 Orelvo-Study Treatment

Company Code:

Chemical Name:

Empirical Formula:

Generic Name: Voclosporin

Dosage Form: Softgel capsules

Strength: 7.9 mg of voclosporin per softgel capsule

Manufacturer:

#### 7.1.2 Placebo Control

Placebo softgel capsules, identical to 7.9 mg Orelvo softgel capsules, will be provided.

#### 7.1.3 Background Therapy

#### 7.1.3.1 Mycophenolate Mofetil

Oral MMF in the form of 500 mg tablets will be centrally supplied by Aurinia. Aurinia will reimburse the cost of the MMF tablets if not centrally provided by Aurinia to the sites.

#### 7.1.3.2 Corticosteroids

Oral corticosteroids will be prescribed at the investigational sites and costs will be reimbursed by Aurinia.

# 7.2 Drug Dosage and Administration

#### 7.2.1 Treatment Arms

Subjects will receive a maximum of either 3 capsules of Orelvo (23.7 mg BID) or matching placebo BID.

Subjects will commence dosing with either oral Orelvo or matching placebo, as randomized into AURORA 1, at the same dose as was given at the time of completion of the AURORA 1 study.

#### Orelvo – 23.7 mg (3 capsules) BID

Orelvo 23.7 mg BID; maximum of 3 capsules administered BID in combination with MMF and oral corticosteroids, if applicable, from consent onwards.

#### Placebo – 3 capsules BID

Placebo; 3 capsules administered BID in combination with MMF and oral corticosteroids from consent onwards.

After 12 months treatment in the AURORA 2 Continuation Study (i.e., 24 months treatment in total), subjects with controlled UPCR (in the Investigator's opinion), taking the 23.7 mg (3 capsules) BID dose will be permitted to reduce the dose of Orelvo to 15.8 mg (2 capsules) BID if considered appropriate and at the discretion of the Investigator and after consultation with the Medical Monitor.

#### 7.2.2 Dosing Guidelines

#### 7.2.2.1 Orelvo/Placebo – Study Treatment

Study treatment will be taken BID with water on an empty stomach as close to a 12 hour schedule as possible, and with a minimum of 8 hours between doses. If the subject misses a dose of study treatment by less than 4 hours from the anticipated dosing time, the missed dose will be taken immediately. The next dose will be taken at the originally scheduled time. If a missed dose of study treatment is greater than 4 hours from the expected dosing time, the subject will skip the dose and take the next dose at the originally scheduled time. The variation in dosing will be recorded in the eCRFs. The dose/doses of study treatment may be held at the discretion of the Investigator. Subjects must avoid consumption of grapefruit or grapefruit-containing juice (e.g., pomelo) for the duration of their participation in the study.

**Possible dose adjustments:** If GI or other disturbances occur with study treatment, then study treatment dosing may be reduced or interrupted, and/or appropriate treatment may be initiated (e.g., addition of a proton pump inhibitor (see Appendix 6) and Section 7.6, Orelvo/Placebo Dose Modification).

All unused study treatments (and any empty containers) dispensed to the subject will be returned at each study visit for capsule counts to check compliance. The Investigator will count the returned study treatment and this information will be used to assess subject compliance.

This study treatment count must be documented in the eCRF and source documentation.

#### 7.2.2.2 Corticosteroids

All subjects will continue to receive oral corticosteroids starting at the same dose as at the end of the AURORA 1 study. When clinically indicated, subjects are allowed to be completely titrated off of oral corticosteroids. The sites will contact the Medical Monitor if the dose of oral corticosteroids is to be increased.

## 7.2.2.3 Mycophenolate Mofetil (Background Therapy)

All subjects will continue to receive background therapy of MMF starting at the same dose as at the end of the AURORA 1 study.

• Subjects must be reminded on the risk of pregnancy while taking MMF and the need for adequate contraceptive precautions (see Section 5.4, Adequate/Effective Contraception).

All subjects will take MMF BID (morning and evening), before meals (i.e., on an empty stomach), with a glass of water. If a dose is missed, the subject should take the next correct dose rather than "doubling up" at the next dosing time point. A stable dose of MMF will be maintained throughout the study. Dose changes or interruptions are permitted for clearly documented safety reasons only.

- The target dose of MMF is 2g/day. MMF administration should continue throughout this continuation study at the same dose as taken at the end of the AURORA 1 study. Approval by the Medical Monitor is required for subjects changing the dose of MMF(e.g., total daily dose of 1 or 3 g/day) from enrolment onwards.
- If GI disturbance or other side-effects occur with MMF, the 1 g BID dosing may be changed to 500 mg four times daily.
- If a subject has an absolute neutrophil count (ANC) <1,500/mm³ at any study visit, the dose of MMF should be decreased or interrupted. If a subject has an ANC <1,000/mm³ at any visit, the dose should be discontinued and only recommenced when the ANC reaches 1,500/mm³. If the subject has a dose interruption of MMF of >14 days, then permanent discontinuation of MMF, therefore the study, should be considered after discussion with the Medical Monitor.
- If deemed necessary by the Investigator on account of leukopenia or other adverse effect, or if the subject weighs 50 kg or less, the dose of MMF may be decreased to a minimum of 500 mg BID.

## 7.3 Package and Labeling

All study treatments provided by Aurinia will be packaged and labeled for Aurinia by appropriately qualified vendors according to all applicable local and country regulatory requirements. All packaging and labeling operations will be performed according to GMP and Good Clinical Practice (GCP).

Study-treatment wallets provided to sites and to subjects will be labeled in the appropriate local language, according to local regulatory requirements.

Wallet label information will be appropriately documented in the Drug Accountability Form after the container has been dispensed to the subject.

## 7.4 Study Treatment Allocation

The IRT system utilized in AURORA 1 will continue to be used for AURORA 2.

## 7.5 Site Supply, Storage, Accountability

## 7.5.1 Site Supply

Once a site has been approved for study initiation, the site will be supplied with an initial stock of study treatment. The need for study treatment resupply will be assessed on a regular basis taking into account the number of subjects enrolled at the site.

# 7.5.2 Storage

Orelvo softgel capsules and matching placebo capsules will be supplied in cartons containing 168 capsules in 4 wallets of 42 capsules each.

The Investigator must ensure the availability of proper storage conditions. All study treatment supplies provided for this study will be stored in a secure area with restricted access at the study site. The capsules must be stored at a controlled room temperature between 15 and 30°C (59-86°F). The Investigator must document and inform the Site Monitor about temperature deviations outside the acceptable range. Subjects will be instructed to store the study treatment at room temperature between 15 and 30°C (59-86°F).

Each site should have a thermometer that records minimum and maximum temperatures daily. Maintenance of a temperature log is mandatory. The log should be updated by site personnel during normal working hours. This log must be available for review by the Site Monitor during on-site monitoring visits.

#### 7.5.3 Accountability

The Investigator at each site is responsible for study treatment supplies. The Investigator will ensure that adequate records of the receipt, dispensing, and return of the study treatment are kept and that the study treatment is used only for subjects enrolled in the study. All data regarding the study treatment must be recorded on the relevant forms provided.

Each study site will maintain a drug inventory/dispensing record for all drugs dispensed and returned. At the end of the study, 1 copy of the drug inventory/dispensing record should be sent to Aurinia for the central study file. The original will be kept in the site files.

After completion of the study, or if it is prematurely terminated, all unused materials will be returned to Aurinia. The decision to destroy study treatment at a site must be made by Aurinia. If the study treatment is destroyed at a site, the Investigator must receive Aurinia approval of the process and forward the certificate of destruction to Aurinia.

Records of oral corticosteroids and MMF must be maintained (prescribed dose, dose adjustments and reasons) in the source notes and must be transcribed into the eCRF.

#### 7.6 Orelvo/Placebo Dose Modification

If GI or other disturbances occur with study treatment, then study treatment dosing may be reduced or interrupted, and/or appropriate treatment may be initiated (e.g., addition of a proton pump inhibitor (see Appendix 6).

After 12 months treatment in the AURORA 2 Continuation Study (i.e., 24 months treatment in total), subjects with controlled UPCR (in the Investigator's opinion), taking the 23.7 mg (3 capsules) BID dose will be permitted to reduce the dose of Orelvo to 15.8 mg (2 capsules) BID if considered appropriate and at the discretion of the Investigator and after consultation with the Medical Monitor.

Where a dose reduction is considered, the following guidance should be considered:

| AURORA 2: Week 52 Dose | AURORA 2: Reduced Dose |
|---------------------------------|------------------------|
| 23.7 mg BID and UPCR ≥1.5 mg/mg | No reduction |
| 23.7 mg BID and UPCR <1.5 mg/mg | 15.8 mg BID |
| <23.7 mg BID | No reduction |

Notes: BID = Twice daily; UPCR = Urine protein creatinine ratio

For any subject receiving an Orelvo (or matching placebo) dose of <23.7 mg BID and presenting with 2 consecutive clinically relevant (in the opinion of the investigator) increases in UPCR, a dose increase of voclosporin (to a maximum of 23.7 mg BID) or appropriate rescue therapy per the Investigator's discretion and current treatment guidelines should be considered.

Dose modifications for background therapy (MMF and corticosteroids) are detailed in Section 7.2, Drug Dosage and Administration.

#### 7.6.1 Deterioration in Renal Function

Serum creatinine and eGFR utilizing the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) formula will be used for the assessment of renal function at every visit (Visits 15-24 and unscheduled visit(s)). Baseline values from the AURORA 1 study will be used in this study.

It is recognized that eGFR may be unreliable at higher values (>100 mL/min/1.73 m<sup>2</sup>). Lupus nephritis subjects with nephrotic range proteinuria frequently have wide fluctuations in serum creatinine (and therefore eGFR) which are not representative of true renal dysfunction. Chronic kidney disease is defined as eGFR <60 mL/min/1.73 m<sup>2</sup> for  $\geq$ 3 months [20], with or without kidney damage.

## 7.6.1.1 Decrease in eGFR >30% and eGFR <60 mL/min/1.73 m<sup>2</sup>

During the treatment period, any subject experiencing a >30% decrease in eGFR from AURORA 1 baseline to <60 mL/min/1.73 m², will have study treatment interrupted until a repeat test can be performed (unscheduled visit to be completed). If the decrease is confirmed and not due to potential contributing factors (e.g., high baseline eGFR, the addition or modification of non-steroidal anti-inflammatory drugs (NSAIDs), angiotensin converting enzyme (ACE) inhibitors, angiotensin II receptor blockers (ARBs), a concurrent state of dehydration, overdosing with study treatment, lupus renal flare, etc.), the case should be discussed with the Medical Monitor, the study treatment should be withheld, and eGFR retested within 48 hours. If the eGFR decrease is not confirmed, the study treatment can be restarted at 2 capsules BID and increased as tolerated with discussion with the Medical Monitor.

#### 7.6.1.2 Decrease in eGFR $\leq$ 30% and eGFR $\leq$ 60 mL/min/1.73 m<sup>2</sup>

During the treatment period, any subject having a  $\leq$ 30% reduction in eGFR from AURORA 1 baseline to <60 mL/min/1.73 m², should have the influence of potential contributing factors (as described in Section 7.6.1.1, Decrease in eGFR >30% and eGFR <60 mL/min/1.73 m²) ruled out and appropriate corrective action taken. Any subject having a >20- $\leq$ 30% reduction compared to baseline in eGFR to <60 mL/min/1.73 m² will have a confirmation measurement done within approximately 2 weeks (at a planned study visit, if any, or an unscheduled visit is to be completed). The subjects will be managed in the most medically appropriate manner in consultation with the Medical Monitor. The management of the decrease in eGFR may include reduction of dose or temporary interruption.

#### 7.6.1.3 Decrease in eGFR ≤20%

During the treatment period, any subject having a  $\leq$ 20% reduction in eGFR from AURORA 1 baseline will be followed by the Investigator.

## 7.6.1.4 Decrease in eGFR >30% and eGFR $\leq$ 90 mL/min/1.73 m<sup>2</sup>

During the treatment period, any subject having a >30% reduction in eGFR from AURORA 1 baseline to ≤90 mL/min/1.73 m², should have the influence of potential contributing factors (as described in Section 7.6.1.1, Decrease in eGFR >30% and eGFR <60 mL/min/1.73 m²) ruled out and a confirmation measurement done within approximately 2 weeks (at a planned study visit, if any, or an unscheduled visit is to be completed). The subjects will be managed in the most medically appropriate manner in consultation with the Medical Monitor.

#### 7.6.1.5 Decrease in eGFR >30% and eGFR >90 mL/min/1.73 m<sup>2</sup>

During the treatment period, any subject having a >30% reduction in eGFR from AURORA 1 baseline to >90 mL/min/1.73 m<sup>2</sup> (i.e., within normal range) should be monitored by the Investigator for further decline in eGFR. Should further eGFR changes occur, the subjects will be managed in the most medically appropriate manner in consultation with the Medical Monitor and the guidance above.

#### 7.6.1.6 Recovery of eGFR

Subjects experiencing a decrease in eGFR with resultant decrease in dose should be reassessed for recovery of renal function. If the repeated eGFR is >80% of AURORA 1 baseline, the dose should be increased by 1 capsule BID and eGFR assessed within 2 weeks.

#### 7.7 Procedures for Overdose

Based on clinical experience with Orelvo, symptomatic treatment of AEs or overdoses is indicated. Treatment for renal dysfunction, hypertension, and infection may include dose reduction or dose discontinuation. Magnesium supplementation may be required for hypomagnesemia. Treatment for GI complaints and biochemical/hematological abnormalities, and all other expected AEs, should be based on symptoms, with care taken to rule out other causes.

# 7.8 Prohibited Therapy and Concomitant Treatment

Any concomitant treatment given for any reason during the course of the study must be recorded in the eCRF and in the subject's source documents, including dosage, start and stop dates, and reason for use.

Any class of medications not mentioned below and with the potential to interfere with evaluation of the study treatment must be discussed and documented with the Medical Monitor.

#### 7.8.1 Prohibited Medications

The same medications prohibited in the AURORA 1 study will be prohibited in this study.

The following medications cannot be taken during the study:

- IV corticosteroids unless approved by the Medical Monitor
- Enteric-coated oral corticosteroids during the study are not allowed. No other use of non-enteric coated oral corticosteroids, other than administration required as per protocol, is allowed
- IV immunoglobulin treatment
- Cyclophosphamide
- Cholestyramine or other drugs that may interfere with enterohepatic recirculation of MMF
- Initiation of new treatment or change in dosage of ARBs and/or ACE inhibitors
- CNIs (e.g., cyclosporine and tacrolimus)
- Immunosuppression biologic agents (e.g., abatacept, belimumab, infliximab, adalimumab, etanercept, or rituximab)
- Vaccines using live organisms, viral or bacterial
- MMF dose other than 2 g/day without prior discussion with the Medical Monitor
- Concomitant therapy with other immunosuppressants after consent, other than MMF administered per protocol
- AZA or mycophenolate sodium
- Ketoconazole or rifampin
- Concomitant use of other CYP3A4/5 inhibitors and inducers should be discussed with the Medical Monitor

Appendix 7 contains a summary of additional treatment and food restrictions.

#### 7.8.2 Allowed Concomitant Medications

These medications are permitted during the study:

- Topical steroids (e.g., nose, scalp, skin, inhaled)
- Antimalarials should be prescribed when clinically indicated
- Herbal supplements can be used with caution and depending on active ingredients

Treatments which may be used as medically indicated, according to the judgment of the Investigator can be found in Appendix 6. Treatments not included in this list may be acceptable in the study; such treatments should be verified with the Medical Monitor prior to use. A summary of treatment and food restrictions can be found in Appendix 7.

#### 7.9 Increased Blood Pressure

For all subjects, the target systolic pressure is  $\leq$ 130 mmHg and the target diastolic pressure is  $\leq$ 80 mmHg. Investigators should use all means possible permitted in the protocol to maintain the BP within these limits. If no further adjustment of antihypertensive therapy is possible, the subject should be discussed with the Medical Monitor.

If on any study day, systolic BP is >165 mmHg or diastolic BP is >105 mmHg and is associated with symptoms of hypertension (i.e., persistent headache, altered mental status, shortness of breath, chest pain consistent with angina pectoris, symptoms of heart failure, evidence of renal insufficiency of new onset, evidence of hypertensive retinal injury [hemorrhages, papilledema]), study treatment should be withheld, the Medical Monitor contacted, and the subject treated as per Investigator local practices and best judgment. The subject will continue with all study visits per the Schedule of Events. Study treatment must not be reintroduced without prior discussion with the Medical Monitor.

# 8. RISKS/PRECAUTIONS

No evidence available at the time of the completion of this study protocol indicated that special warnings or precautions are required, other than those noted in the IB.

If additional special warnings or precautions become apparent before study completion, Aurinia will notify the Investigator at each site.

## 9. STUDY PROCEDURES

## 9.1 Description of Study Assessments

## 9.1.1 Laboratory Assessments

Analysis of all samples for hematology, chemistry, hepatic function, lipid profiles, proteinuria, and urinalysis will be performed at a central laboratory using standard validated methods (see the laboratory manual). All study data analyses involving laboratory values will be based on results from the central laboratory.

The UPCR will be calculated both from the FMV and from standard urinalysis results. If the FMV is for some reason not available, then standard urinalysis from a 24-hour urine collection may be substituted as an exception but only after agreement is reached with the Medical Monitor.

Blood and urine samples for the following efficacy and safety assessments (See Table 1) will be drawn in accordance with the Schedule of Events.

**Table 1** Review of Laboratory Assessments

| Test Type | <b>Test Parameters</b> | <b>Collection at Visits</b> |
|---|---|---|
| Hematology | Complete blood count (CBC) | All visits |
| | Hematocrit | |
| | Hemoglobin | |
| | Mean corpuscular hemoglobin (MCH) | |
| | Mean corpuscular hemoglobin concentration (MCHC) | |
| | Mean corpuscular volume (MCV) | |
| | Platelet count | |
| | Red blood cells (RBC) | |
| | Red blood cell morphology | |
| | White blood cells (WBC) | |
| | Differential (absolute and %) | All visits |
| | Bands | |
| | Basophils | |
| | Eosinophils | |
| | Lymphocytes | |
| | Monocytes | |
| | Neutrophils | |

Table 1 Review of Laboratory Assessments (Cont'd)

| Test Type | Test Parameters | Collection at Visits |
|---|---|---|
| Blood Chemistry | Alanine aminotransferase (ALT) | All visits |
| | Albumin | All visits |
| | Alkaline phosphatase (ALP) | All visits |
| | Aspartate aminotransferase (AST) | All visits |
| | Bicarbonate | All visits |
| | Bilirubin (direct and total) | All visits |
| | Blood urea nitrogen (BUN) | All visits |
| | Calcium | All visits |
| | Chloride | All visits |
| | Cholesterol (total, HDL, and | Month 24 and Month 36 |
| | LDL) | Every 6 months |
| | Creatine kinase | All visits |
| | Creatinine | All visits |
| | Gamma-glutamyl transferase | All visits |
| | (GGT) | Annually |
| | Glucose | All visits |
| | Glycosolated hemoglobin | All visits |
| | (HbA1c) | All visits |
| | Lactic dehydrogenase (LDH) | All visits |
| | Magnesium | All visits |
| | Phosphorous, inorganic | All visits |
| | Potassium | Annually |
| | Protein, total | All visits |
| | Sodium | |
| | Triglycerides | |
| | C-reactive Protein | |
| Urinalysis | Complete urinalysis (to include urine protein, creatinine, blood, urine microscopy). | All visits |
| Proteinuria | FMV will be performed to analyze UPCR. A 24-hour urine may be substituted for FMV if required. | All visits |
| | FMV | All visits |
| | 24-hour urine | Every 6 months |

Table 1 Review of Laboratory Assessments (Cont'd)

| Test Type | Test Parameters | Collection at Visits |
|---|---|---|
| Pregnancy Test | A serum pregnancy test will be performed for females of childbearing potential. Urine pregnancy tests will be done using a dipstick. | iles of Month 36 (Serum) itial. Urine Month 12, Month 15, Month 18, |
| Lupus Markers | Anti-double-stranded DNA (anti-dsDNA) antibodies | All visits |
| | Serum Complement 3 Complement 4 | All visits |
| Special Tests | Estimated glomerular filtration rate (eGFR) | All visits |

Notes: FMV = first morning void; HDL = High-density lipoprotein; LDL = Low-density lipoprotein; UPCR = urine protein creatinine

Baseline values from the AURORA 1 study will be used in this study.

The total amount of blood that will be collected during the study from an individual subject is approximately 200 mL over 2 years.

For details on whether laboratory abnormalities should be reported as AEs and on the follow-up required in such cases, see Section 10.2.5, Clinical Laboratory Evaluations.

#### 9.1.1.1

#### 9.1.2 Physical Examinations

Physical examinations will be performed in accordance with the Schedule of Events.

The physical examination will include a review of SLE-related manifestations which will also be recorded. An abbreviated physical examination will be conducted at Month 12 from the results of the Week 52/ End of Treatment Visit in the AURORA 1 study, and at Month 36 End of Study or Early Termination as per the Schedule of Events.

The abbreviated examination will consist of checking the normality or abnormality of the following body systems: general appearance, cardiovascular system, and pulmonary system. Any abnormalities will be recorded in the eCRF and reported as an AE. Because the investigational medication is an immunosuppressant, physical examination will include clinical examination for tumors.

Subject weight will also be recorded at each physical examination; however, height is not required.

#### 9.1.3 Vital Signs

The following vital signs will be measured at all visits in accordance with the Schedule of Events:

- Resting BP (systolic and diastolic)
- Resting HR
- Body temperature (°C or °F)

To avoid variability, the same method of obtaining body temperature should be used throughout the study.

#### 9.1.3.1 Blood Pressure Management

BP and heart rate (HR) will be measured with the subject in a sitting position after 5 minutes of rest. The procedure for standardized measurement of BP is detailed in Appendix 2.

If the BP measure is confirmed to be >130/80 mmHg (i.e., by the mean of the second and third repeats of 3 readings), the subject's BP will be managed per local practice. If the BP remains uncontrolled with the maximal doses of first and secondline- antihypertensive therapies referenced in Appendix 1, then the Investigator should contact the Medical Monitor to consider dose adjustment of the study treatment. See Section 7.9, Increased Blood Pressure for management of increased BP.

#### 9.1.4 Standard 12-lead Electrocardiogram

The electrocardiogram (ECG) will be a standard 12-lead tracing performed at the investigational site, assessed by a qualified physician at the investigational site, and retained as a source document. Any abnormalities will be recorded in the eCRF. ECGs will be recorded after the subject has been in a resting, supine position for at least 5 minutes. Abnormal ECG tracings can be reviewed by the Medical Monitor. Significant abnormalities, including findings that may prompt discontinuation of study treatment, must be discussed with the Medical Monitor.

ECGs will be measured at Month 12 from the results of the Week 52/ End of Treatment Visit in the AURORA 1 study, and at Month 18, 24, and 36/End of Study or Early Termination as per the Schedule of Events.

#### 9.1.4.1 Procedures to Manage a Treatment-Emergent Increase in QTc

In the event that a subject has a QT interval duration corrected for heart rate using method of Fridericia (QTcF) value exceeding 500 msec, or an increase >60 msec from AURORA 1 baseline, the Medical Monitor must be informed. The subject will be asked to return for an unscheduled visit within 24 hours and the ECG will be repeated (confirmed), in triplicate (i.e., three 10-second ECGs in rapid succession within 1 minute). If the repeat measurements confirm that the QTcF is >500 msec or >60 msec from baseline, the subject will be withdrawn from treatment with the study treatment and followed until the QTcF value either returns to baseline (or as appropriate) or until, in the judgment of the Investigator, further evaluation is not clinically indicated; study treatment will not be restarted.

If study treatment is discontinued, the subject should continue in the study for all remaining scheduled study visits.

## 9.1.5 Lupus Disease Activity Assessments

The Safety of Estrogens in Lupus Erythematosus National Assessment (SELENA)- Systemic Lupus Erythematosus Disease Activity Index (SLEDAI) assesses disease activity within the last 10 days. Twenty-four items are scored for 9 organ systems, and summed to a maximum of 105 points. A score of 6 is considered clinically significant. See Appendix 5.

Assessments for SELENA-SLEDAI will be conducted at Month 12 from the results of the Week 52/ End of Treatment Visit in the AURORA 1 study, and at Months 18, 24, and 36/End of Study or Early Termination.

## 9.1.6 Kidney Biopsy

At sites that are able to meet the biopsy requirements,

#### 9.2 Schedule of Assessments

A detailed schedule of assessments (including all protocol-required assessments, visits, and visit windows) is located on the Schedule of Events. No study related assessments will be performed (including changes to current medications to meet study eligibility) until the subject has provided signed and dated informed consent. Every effort will be made to keep the subject within the requested visit schedule. If a subject is seen outside of the visit window listed on the Schedule of Events, the reason must be clearly documented in the source notes. The

Investigator (or designee) should contact Aurinia for assistance with getting the subject's schedule back on track in order to avoid large variances in treatment exposure or to avoid delaying overall study timelines.

## **9.2.1 Screening Visit Procedures**

Screening will take place in the AURORA 1 study. In this continuation study, subjects who have completed 52 weeks of treatment with study drug in the AURORA 1 study and have provided signed and dated informed consent will be entered into this study.

Month 12 refers to Week 52/ End of Treatment Visit of the AURORA 1 study.

#### 9.2.2 Treatment Procedures

Subjects who satisfy all of the inclusion and exclusion criteria will be eligible for consent into the AURORA 2 study.

Month 12 refers to Week 52/ End of Treatment Visit of the AURORA 1 study. All subjects will continue to receive background therapy of MMF and oral corticosteroids, if applicable, starting at the same dose as at the end of the AURORA 1 study. When clinically indicated, subjects are allowed to be completely titrated off of oral corticosteroids; the sites will contact the Medical Monitor if the dose of oral corticosteroids is to be increased. Subjects will be fasting for 8 hours on the day of study entry on Month 12 (Week 52/ End of Treatment Visit of the AURORA 1 study), at Month 24, and at Month 36 End of Study visit.

Subjects will complete all assessments per the Schedule of Events at Month 12 and at Months 15, 18, 21, 24, 27, 30, and 33. Subjects will continue to receive either Orelvo or matching placebo as randomized in the AURORA 1 study at appropriate visits.

Adverse events and concomitant medication will be recorded prior to the conduct of other study assessments at each visit.

Assessments at visits during the treatment period include:

- HRQoL (SF-36) will be answered by and collected from the subject, as first study procedure, at Month 12, provided from the results of Week 52/ End of Treatment Visit of the AURORA 1 study, and at Months 18, 24, and 30.
- Abbreviated physical examination (including body weight) at Month 12, provided from the results of Week 52/ End of Treatment Visit of the AURORA 1 study.
- Vital signs (BP, pulse, temperature) at all visits; Month 12 assessments will be provided from the results of Week 52/ End of Treatment Visit of the AURORA 1 study.

- Standard 12-lead ECG at Month 12, provided from the results of Week 52/ End of Treatment Visit of the AURORA 1 study, and at Months 18 and 24.
- Blood and urine sample collection for analysis at central laboratory at all visits; Month 12 assessments will be provided from the results of Week 52/ End of Treatment Visit of the AURORA 1 study.
- FMV urine sample collection at all visits; Month 12 assessments will be provided from the results of Week 52/ End of Treatment Visit of the AURORA 1 study.
- 24-hour urine collection at Month 12, provided from the results of Week 52/ End of Treatment Visit of the AURORA 1 study, and at Months 18, 24, and 30 (IMPORTANT: 24-hour urine collection will have to begin 2 days prior to the scheduled visit in order not to coincide with the FMV sampling due on the day of this visit).
- Pregnancy testing and immunology at all visits; serum pregnancy testing at Month 12 and Month 24 and urine pregnancy testing at Month 12, Month 15, Month 18, Month 21, Month 27, Month 30, and Month 33.
- AEs at all visits; Month 12 assessments will be provided from the results of Week 52/ End of Treatment Visit of the AURORA 1 study.
- Concomitant medications at all visits; Month 12 assessments will be provided from the results of Week 52/ End of Treatment Visit of the AURORA 1 study.
- SELENA-SLEDAI will be evaluated at Month 12, provided from the results of Week 52/ End of Treatment Visit of the AURORA 1 study, and at Months 18 and 24.
- Study treatment dispensing (including study treatment and background therapy) at all visits.
- Returned capsule count and drug accountability at all visits.
- Information for the HRU assessment will be collected and recorded at all visits; Month 12 assessments will be provided from the results of Week 52/ End of Treatment Visit of the AURORA 1 study.

## 9.2.3 End of Study (or Early Discontinuation) Procedures

On completion of treatment at Month 36 or earlier if subject is discontinued/withdrawn early, all assessments for Visit 23 (End of Study or Early Termination) will be completed per the Schedule of Events. See also Section 5.5, Withdrawal of Subjects, for further information on withdrawal procedures and criteria.

The following assessments for the end of study visit will be performed:

- SF-36
- Abbreviated physical examination (including body weight)
- Vital signs (BP, pulse, temperature)
- Standard 12-lead ECG
- Blood sample collection for analysis at central laboratory
- Serum pregnancy testing
- FMV
- 24-hour urine sample collection (IMPORTANT: 24-hour urine collection will have to begin 2 days prior to Month 36 visit in order not to coincide with the FMV sampling due on the day of this visit)
- Concomitant medication
- AEs
- SELENA-SLEDAI
- Returned capsule count and drug accountability
- Confirmation of completion/discontinuation using IRT
- Information for the HRU assessment will be collected and recorded

## 9.2.4 Follow-up Procedures

All subjects will have a safety follow-up visit after the last dose of study drug at Month 37 ( $\pm 10$  days), to collect any new AEs and concomitant medications. This visit (Visit 24) will be

conducted as an in-clinic visit. An assessment of vital status will also be conducted at 6 and 12 months post study.

Assessments for the follow-up visit are as follows:

- Vital signs (BP, pulse, temperature)
- Blood sample collection for analysis at central laboratory (eGFR)
- FMV urine sample collection
- Concomitant medication
- AEs
- Confirmation of completed follow-up visit using IRT
- Assessment of vital status will occur at 6 and 12 months post study

#### 9.2.5 Unscheduled Visit

Unscheduled visits may be performed during the course of the study for safety reasons. An unscheduled visit is required 2 weeks after dose reduction at any time during the study. Only the data relevant to the purpose of the visit will be collected in the source documents and eCRF. An unscheduled visit is requested in the following cases:

- QTcF value exceeding 500 msec, or an increase >60 msec from baseline, where the ECG will be repeated (confirmed) at an unscheduled visit
- Systolic BP is ≥165 mmHg or diastolic BP is ≥105 mmHg, or confirmed systolic BP >130 mmHg or a diastolic BP >80 mmHg
- Decrease in eGFR >30% compared to baseline, or a confirmed decrease in eGFR >20-30% compared to baseline (detailed in Section 7.6.1, Deterioration in Renal Function)

Additional unscheduled visits may be planned per Investigator's judgment.

## 9.3 Study Specific Assessment Procedures

## 9.3.1 Health-related Quality of Life Assessments (HRQoL)

## 9.3.1.1 Short Form Health Survey (SF-36)

The SF-36 HRQoL assessment is a 36-question subject HRQoL questionnaire and is presented in Appendix 8.

## 9.3.2 Healthcare Resource Utilization (HRU) Assessment

The collection of information on HRU will be collected at the time points specified in the Schedule of Events (Month 12, provided from the results of Week 52/ End of Treatment Visit of the AURORA 1 study, and at Months 15, 18, 21, 24, 27, 30, 33, and 36) and documented in the electronic data capture (EDC) system. This information will be collected via interview of the subject by the study staff and entered into the EDC system. General information collected may include:

- Type of insurance coverage
- Number of visits to ANY health care professionals (HCP), other than study doctor
- Types of HCP visited (specialists versus primary care)
- Time spent on visits
- Diagnostic tests performed
- Time spent by caregivers assisting patient with HCP visits (can ask general question if subject required a family member or other person to assist them to attend the visit)
- Prescriptions issued, filled
- Community services used

# 10. EVALUATION, RECORDING AND REPORTING OF AES AND SAES

#### 10.1 Definitions

#### 10.1.1 Adverse Event

Any untoward medical occurrence in a subject administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment is an AE. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product.

## 10.1.2 Adverse Drug Reaction

In the pre-approval clinical experience with a new medical product or its new usages, particularly as the therapeutic dose(s) may not be established, all unintended responses to a medicinal product related to any dose should be considered adverse drug reactions (ADRs). The phrase "responses to a medicinal product" means that a causal relationship between a medicinal product and an AE is at least a reasonable possibility, i.e., the relationship cannot be ruled out.

#### 10.1.3 Serious Adverse Event

An SAE (experience) or reaction is an untoward medical occurrence that at any dose meets 1 or more of the following criteria:

- Results in death (Note: death is an outcome, not an event)
- Is life-threatening (Note: the term "life-threatening" refers to an event in which the subject was at immediate risk of death at the time of the event; it does not refer to an event which could hypothetically have caused a death had it been more severe)
- Requires in-patient hospitalization or prolongation of existing hospitalization
- Results in persistent or significant disability/incapacity
- Results in a congenital anomaly/birth defect
- Is a medically important event or reaction

The definitions and reporting requirements of International Council for Harmonisation (ICH) Guidelines for Clinical Safety Data Management, Definitions, and Standards for Expedited Reporting, Topic E2 will be adhered to.

Medical and scientific judgment must be exercised in deciding whether expedited reporting is appropriate in other situations, such as important medical events that may not be immediately life-threatening or result in death or hospitalization but may jeopardize the subject or may require intervention to prevent one of the other outcomes listed in the definition above. These will also usually be considered serious.

Hospitalizations for elective or previously scheduled surgery for pre-existing conditions, which have not worsened after initiation of treatment, will not be classed as SAEs. Previously scheduled hospitalizations must be documented in the subject's source documents before the subject signed the informed consent form (ICF). A kidney biopsy performed as part of the study to verify eligibility will not be considered an SAE. Any complication experienced during a kidney biopsy procedure resulting in hospitalization or a prolongation of the hospitalization requires SAE reporting.

## 10.1.4 Suspected Unexpected Serious Adverse Reaction

Any ADR that is both serious and unexpected (per the IB) that, based on the opinion of the Investigator or Aurinia, is felt to have a reasonable suspected causal relationship to a medicinal product is a suspected unexpected serious adverse reaction.

## **10.2** Adverse Event Descriptors

## 10.2.1 Intensity/Severity Categorization

The term "severe" is often used to describe the intensity (severity) of a specific event (as in mild, moderate, or severe myocardial infarction); however, the event itself may be of relatively minor medical significance (such as severe headache). This is not the same as "serious," which is based on subject/event outcome or action criteria usually associated with events that pose a threat to a subject's life or functioning. Seriousness (not severity) serves as a guide for defining regulatory reporting obligations.

In general, the intensity of a particular AE to be recorded is the worst intensity experienced by the subject during the course of the event. The medical assessment of intensity will be determined by using the following definitions:

Mild: The AE is easily tolerated and does not interfere with usual activity.

Moderate: The AE interferes with daily activity, but the subject is still able to function.

Severe: The AE is incapacitating and the subject is unable to work or complete usual

activity.

## 10.2.2 Causal Relationship Categorization

An Investigator who is qualified in medicine must make the determination of relationship to the study treatment for each AE and SAE. The Investigator must decide whether, in his or her medical judgment, there is a reasonable possibility that the event may have been caused by the study treatment. If there is no valid reason for suggesting a relationship, then the AE/SAE must be classified as not related. Otherwise, if there is any valid reason, even if undetermined or untested, for suspecting a cause-and-effect relationship between the study treatment and the occurrence of the AE/SAE, then the AE/SAE will be considered related. For SAEs, the Investigator must provide a brief comment explaining the rationale of his/her assessment of causal relationship on the SAE reporting form.

The following additional guidance may be helpful:

| Term | Relationship | Definition |
|---|---|---|
| Related | Yes | The temporal relationship of the clinical event to study drug administration indicates a causal relationship, and other drugs, therapeutic interventions or underlying conditions do not provide a sufficient explanation for the observed event. |
| Not related | No | The temporal relationship of the clinical event to study drug administration does not indicate a causal relationship, or other drugs, therapeutic interventions or underlying conditions provide a sufficient explanation for the observed event. |

If the causal relationship between an AE/SAE and the study treatment is determined to be "related", the event will be considered to be related to study treatment for the purposes of expedited regulatory reporting. In circumstances where the Investigator has not yet provided his/her assessment about the relationship, the event will be considered as "related" and qualify for expedited regulatory reporting.

## **10.2.3 Outcome Categorization**

Outcome may be classified as recovered without sequelae; recovered with sequelae; improved; worsened; ongoing; ongoing at End of Study; fatal; or unknown. If the outcome is reported as recovered with sequelae for an SAE, the Investigator should specify the kind of sequelae on the SAE reporting form. SAEs that are ongoing at the time of death will have an outcome of "unknown" recorded. SAEs resulting in a fatal outcome will have an outcome of "fatal" recorded.

## 10.2.4 Symptoms of the Disease Under Study

Symptoms and fluctuations in laboratory parameters related to the disease under study will not be classed as AEs as long as they are within the normal day-to-day fluctuation of the disease. An explanation of these circumstances must be written in the source documents.

Worsening of the symptoms or laboratory parameters however, will be recorded as an AE, and clearly marked as worsening or by the subject's worst observed intensity. The Investigator will be required to assess the relationship to disease under study for each AE as related or not related. An AE will not be able to be assessed as related to both disease under study and related to study treatment.

## 10.2.5 Clinical Laboratory Evaluations

A change in the value of a safety laboratory investigation can represent an AE if the change is clinically relevant in the opinion of the Investigator or if, during treatment with the study treatment, a shift of a parameter is observed from a normal value to a pathological value, or a further worsening of an already pathological value.

If, at the end of the treatment phase, there are pathological laboratory values which were not present at baseline, further clinical or laboratory investigations will be performed until the values return to within reference range or until a plausible explanation (e.g., concomitant disease) is found for the pathological laboratory values.

If the Investigator considers such an AE as serious it must be reported as an SAE.

#### 10.2.6 Abuse, Misuse, Overdose and Medication Error

All AEs of special interest such as study treatment abuse, misuse, overdose, and medication error have to be documented in the subject's eCRF and source documentation. If any occurrence of abuse, misuse, overdose, or medication errors leads to any event that fulfils any seriousness criteria, the event has to be reported as an SAE.

# 10.3 Reporting Procedure for AEs, SAEs, and Pregnancy

#### **10.3.1 Adverse Events**

All AEs either observed by the Investigator or one of his/her medical collaborators, or reported by the subject spontaneously, or in response to a direct question, will be noted in the AE section of the subject's eCRF and source documentation. This applies to all AEs regardless of presumed relationship to the study treatment. Adverse events leading to discontinuation of study treatment must be collected.

If any AE is reported, the date of onset, relationship to disease under study, relationship to study treatment, any action taken, date of resolution (or the fact that it is still continuing or has become chronic), outcome, and whether the AE is serious or not, will be recorded. Use of colloquialisms and abbreviations should be avoided. Only 1 AE term should be recorded in the event field on the AE eCRF. Where possible, the Investigator should report a diagnosis rather than signs and symptoms or abnormal laboratory values. However, if a constellation of signs and/or symptoms cannot be medically characterized as a single diagnosis or syndrome at the

time of reporting, each individual event should be recorded on the AE eCRF. If a diagnosis is subsequently established, all previously reported AEs based on signs and symptoms should be nullified by the Investigator and replaced by one AE report based on the single diagnosis, with a starting date that corresponds to the starting date of the first symptom of the eventual diagnosis.

The AE reporting period begins at the time the ICF is signed by the subject. The AE reporting period ends at the study follow-up visit (Visit 24). Adverse events persisting at the time of study completion will be followed by the Investigator through contact with the subject until resolution or stabilization has occurred (or the subject is lost to follow-up and cannot be contacted) and recorded in the source documents. If the subject reports an AE, it is the Investigator's responsibility to acquire sufficient information in order to assess causality. This may require additional laboratory testing, physical examinations, telephone contacts, etc. In circumstances where the Investigator is unable to make contact with the subject, the Investigator must provide a written statement to Aurinia confirming that the subject is lost to follow-up.

In order to avoid bias in eliciting AEs, subjects should be asked a non-leading question, such as "How are you feeling?" It is also important to question the subject in a non-leading way about changes in their health or concomitant medication usage since their last visit. This information should be collected prior to completion of assessments at all study visits. In addition, any symptoms/conditions reported during assessments and deemed to be clinically significant by the Investigator will be considered AEs.

#### 10.3.2 Serious Adverse Events

All SAEs occurring after the signing of the ICF will be reported to within 24 hours of the Investigator, designee, or site staff's knowledge of the event regardless of relationship to study treatment or relationship to disease under study. All SAEs are to be reported on the eCRFs.

In the event that the site experiences a temporary disruption of the EDC system a back-up paper SAE Reporting Form will be available for site staff to complete.

- Site staff will complete the paper SAE report form and e-mail it within 24 hours to the following address:
- Only in cases where the email system is unavailable, site staff will send the SAE by fax to: (US) and (Outside US).

If notification is made via email or fax, site staff must enter the SAE information into the EDC system as soon as the system becomes available.

All SAEs, regardless of causality, will be reported from the time the ICF is signed until 30 days following the last study visit or 30 days after last study treatment administration in subjects who withdraw or discontinue prior to study completion. No formal study visit is required but Investigators must report any SAEs that occur during this 30 day period on the eCRF. If the Investigator has not seen the subject at a clinic visit at the end of the reporting period, the Investigator must make reasonable efforts to contact the subject to inquire about SAEs.

All recorded SAEs, regardless of relationship to disease under study or relationship to study treatment, will be followed up until resolution, stabilization, or the subject is lost to follow-up and cannot be contacted. In circumstances where the Investigator is unable to make contact with the subject, the Investigator must provide a written statement to Aurinia confirming that the subject is lost to follow-up.

Any SAE considered to have a causal relationship (i.e., "related") to the study treatment and discovered by the Investigator at any time after the study will be reported. A rationale for the assessment of a causal relationship must be provided by the Investigator. The Investigator will also be required to assess the relationship to disease under study for each SAE as related or not related. An SAE will not be able to be assessed as related to both disease under study and related to study treatment. Any safety information that is obtained after the Follow-up Visit (Visit 24) will be documented in the safety database only.

A death occurring during the study or which comes to the attention of the Investigator within 30 days after the last study visit (including the Follow-up Visit) or until 30 days after the last study treatment administration, whichever is longer, whether considered treatmentrelated or not, must be reported to Aurinia-. If the subject died, the SAE report should include the cause of death as the event term and whether or not the death was related to study treatment, as well as the autopsy findings, if available. Preliminary reports will be followed by detailed descriptions which will include copies of hospital case reports, autopsy reports/certificates and other documents when requested and applicable.

Additional follow-up information must be reported in the eCRF within 24 hours of awareness following Investigator (or site) awareness of the information. The Investigator should not delay reporting an SAE in order to obtain additional information. Additional information, when available, should be reported to by the reporting procedures described above.

The Investigator is encouraged to discuss with the study Medical Monitor when the issue of seriousness is unclear or questionable.

An Investigator who receives an Investigator safety report describing an SAE or other specific safety information (e.g., summary or listing of SAE) from the sponsor will file it along with the IB and will notify the IRB/IEC, if appropriate according to local requirements.

The sponsor or its representative will be responsible for determining and, in turn, reporting SAEs to regulatory authorities according to the applicable regulatory requirements.

## 10.3.3 Pregnancy

Pregnancy occurring in a female subject or in the partner of a male subject should be reported to within 24 hours of becoming aware of the event using the pregnancy eCRF. The Investigator should counsel the subject, and in the case of a male subject, the subject's partner, discuss the risks of continuing with the pregnancy and the possible effects on the fetus. A female subject must immediately inform the Investigator if she becomes pregnant during the study. Monitoring of the pregnancy in a female subject should continue until conclusion of the pregnancy. In case of a pregnancy in the partner of a male subject, the Investigator should obtain informed consent of the pregnant partner prior to monitoring of the pregnancy.

Women who have a positive pregnancy test during the study will be withdrawn from the study treatment and the procedures for withdrawal will be completed. The Medical Monitor must be contacted immediately to break the blind (if applicable).

All pregnancies, subject or partner of a subject, that occur during the study or come to the attention of the Investigator within 30 days after the last study visit (including the Follow-up Visit) or until 30 days after last study treatment administration, whichever is longer, must be reported to by the reporting procedures described above.

The outcome of all such pregnancies (including normal births) should be followed up and documented, even if the subject was withdrawn from the study. Every effort should be made to gather information regarding the pregnancy outcome until 90 days (or otherwise as appropriate) post-partum. It will be the responsibility of Aurinia, together with the appropriate support of the Investigator, to obtain this information.

Complications of pregnancy such as abortion (spontaneous or induced), premature birth, or congenital abnormality are considered SAEs and should be reported following the reporting procedures as outlined in Section 10.3.2, Serious Adverse Events. In the event that the site experiences a temporary disruption of the EDC system, a back-up paper Pregnancy Reporting Form will be available for site staff to complete.

# 11. CLINICAL ENDPOINTS COMMITTEE

A CEC will be constituted to adjudicate the following secondary endpoints for subjects in this study:

- Renal flare
- Extra-renal flare

The CEC will adjudicate the endpoints by reviewing blinded data. Aurinia will establish a charter document explaining the working procedures and responsibilities of the CEC. All adjudication decisions of the CEC will be appropriately documented.

#### 12. DATA AND SAFETY MONITORING BOARD PROCEDURES

A DSMB will be constituted to protect the safety of study participants. The DSMB will receive blinded eCRF data in the form of tables and listings (prepared by an independent statistician), and review subject status changes and dosing decisions (where appropriate). Where appropriate, the DSMB may receive unblinded data (on a subject level or treatment group level) that should be reviewed in a closed session. Examples of the data that may be included are: disposition, demographics, baseline characteristics, AE data, SAE data (by severity and causality), laboratory data, dose adjustments, protocol adherence, and subject withdrawals. The DSMB will evaluate the progress of the study, assess data quality and timeliness, participant recruitment, accrual and retention, and participant benefit versus risk. In addition, the DSMB will monitor external factors relevant to the study, for example scientific and therapeutic developments that may affect participant safety or ethical status. Based on the observed benefits or adverse effects, the DSMB will make recommendations to Aurinia concerning continuation, termination, or modifications of the study.

Aurinia will establish a charter document explaining the working procedures and responsibilities of the DSMB. All deliberations and decisions of the DSMB will be appropriately documented.

## 13. STATISTICAL ANALYSIS

#### 13.1 Statistical Methods

Complete details of the statistical and analytical methods will be provided in a formal Statistical Analysis Plan (SAP), which will be finalized prior to the database lock. A general description of the planned methods is provided below. Any deviation from the SAP will be noted and explained in the clinical study report.

## 13.2 Sample Size and Power Calculations

Subjects will enter this protocol from the AURORA 1 study in order to provide the opportunity of an additional 24 months of treatment (total of 36 months of treatment); no sample size calculation is required.

## 13.3 Populations

#### 13.3.1 Intent-to-Treat Set

The intent-to-treat (ITT) set will be based on ITT principles and will consist of all subjects who are consented to treatment. This group will be analyzed based on the treatment to which the subject was randomized in the AURORA 1 study.

## 13.3.2 Safety Set

The safety set will consist of all subjects who receive at least 1 dose of study drug in the continuation study. The subjects in this group will be analyzed based on the treatment they received. Subjects who receive treatment from more than 1 arm will be assigned to the Orelvo arm.

# 13.4 Background and Demographic Characteristics

Demographic and clinical disease characteristics will be summarized by treatment arm in a descriptive manner but no statistical tests will be performed.

# 13.5 Study Treatment

Compliance to the study treatment will be determined by dividing the number of softgel capsules taken by the expected number of softgel capsules to be taken (based on prescribed dose) over the subject's participation in the study.

Results will be summarized by means of descriptive statistics (n, mean, standard deviation, median, minimum, and maximum) and frequency tables, by treatment arm.
## 13.6 Concomitant Therapy

All concomitant medications will be coded by the WHO Anatomical Therapeutic Chemical Drug Reference List classification. The version used will be provided in the clinical study report.

## 13.7 Endpoint Evaluations

## 13.7.1 Primary Safety Endpoint

The primary safety endpoint is as follows:

• AE profile and routine biochemical and hematological assessments

## 13.7.2 Secondary Efficacy Endpoints

## 13.7.2.1 Key Secondary Efficacy Endpoints

- Proportion of subjects in renal response at Months 12, 18, 24, 30, and 36 defined as:
  - UPCR of  $\leq 0.5$  mg/mg
  - eGFR ≥60 mL/min/1.73 m<sup>2</sup> or no confirmed decrease from baseline in eGFR of >20%
  - Received no rescue medication for LN (see Section 7.8, Prohibited Therapy and Concomitant Treatment)
  - Did not receive more than 10 mg prednisone for ≥3 consecutive days or for
     ≥7 days in total during the 8 weeks prior to the renal response assessment
- Subjects who withdraw from the study prior to the response assessment will be defined as non-responders.
- Proportion of subjects in partial renal response at Months 12, 18, 24, 30, and 36 defined as a 50% reduction from baseline in UPCR.
- Renal flare as adjudicated by the CEC.
- Extra-renal flare as adjudicated by the CEC.
- SELENA-SLEDAI scores by visit.
- Change in UPCR, eGFR, urine protein, and serum creatinine from AURORA 1 baseline.

#### 13.7.2.2 Other Secondary Efficacy Endpoints

- Change in immunology parameters (C3, C4, and anti-dsDNA) from AURORA 1 baseline.
- Change in HRQoL (SF-36) from AURORA 1 baseline.
- HRU.

13.7.2.3

## 13.8 Statistical and Analytical Methods

## 13.8.1 Safety Analysis

The primary safety endpoints are the AE profile and routine biochemical and hematological assessments at Month 36 (Section 13.7.1, Primary Safety Endpoint).

## 13.8.2 Efficacy Analysis

All the secondary efficacy analyses will be performed on the ITT set. Data for each visit (as well as change from AURORA 1 study baseline as required) will be summarized by treatment group and visit for each secondary endpoint.

#### 13.8.2.1 Response Endpoints

The following key secondary efficacy endpoints will be analyzed using the ITT population using logistic regression with terms for treatment group, baseline UPCR, biopsy class, and MMF use at baseline (from AURORA 1) in the model.

- Proportion of subjects in renal response at Months 12, 18, 24, 30, and 36.
- Proportion of subjects in partial renal response at Months 12, 18, 24, 30, and 36.

The results will be expressed as an odds ratio (and associated two-sided 95% CI) for Orelvo compared to placebo. Odds ratios greater than unity show the odds of response are greater for Orelvo than for placebo and therefore indicate a benefit of the Orelvo treatment arm.

#### 13.8.2.2 Renal flare and Extra-renal flare

The proportion of subjects with renal and extra-renal flares (as adjudicated by the CEC) will be analyzed in a similar fashion to the proportion of subjects achieving response.

#### 13.8.2.3 Change from Baseline Endpoints

The following secondary endpoints will be analyzed using a Mixed Effect Model Repeated Measures (MMRM). The MMRM model will include terms for treatment, visit, treatment by visit interaction, and baseline. Results will be expressed as differences between treatment arms (along with the associated 95% CI).

- Change in UPCR, eGFR, urine protein, and serum creatinine from AURORA 1 baseline at each visit.
- Change in immunology parameters (C3, C4, and anti-dsDNA) from AURORA 1 baseline at each visit.
- Change in HRQoL (SF-36) from AURORA 1 baseline at Months 12, 18, 24, 30, and 36.
- Change in SELENA-SLEDAI scores by visit at Months 12, 18, 24, and 36.

## 13.8.2.4 Healthcare Resource Utilization (HRU)

• Healthcare Resource Utilization at Months 12, 15, 18, 21, 24, 27, 30, 33, and 36. Key aspects will be summarized by visit and changes over time will be explored.

## 13.9 Safety Evaluations

Specific safety endpoints are as follows:

- Biochemical (including liver function tests) and hematological laboratory tests
- AE profile and routine biochemical and hematological safety parameters
- Vital signs (BP, HR, temperature) at specific time points and change from baseline
- Standard 12-lead ECGs change from baseline
- Discontinuations from treatment
- Concomitant medications

Laboratory values, vital signs, and other safety parameters providing numeric data will be summarized by visit as absolute values and change from baseline. Laboratory values outside of defined normal ranges will be summarized.

Adverse events will be coded using the latest available version of the Medical Dictionary for Regulatory Activities, the version of which will be provided in the clinical study report.

Treatment-emergent adverse events will be summarized by treatment arm, system organ class, and preferred term. SAEs, SAEs that led to death, and SAEs/AEs that led to withdrawal will also be summarized and listed.

Only AEs which started on or after the date of first dose of study treatment in AURORA 2 will be considered TEAEs, though all AEs after informed consent will be recorded. SAEs occurring at any time after informed consent will be summarized. All concomitant medications will be summarized.

Details of these and other analyses will be provided in the SAP.

All study data analyses involving laboratory values will be based on results from the central laboratory.

## 13.10 Interim Analyses

The study will incorporate an unblinded, interim analysis of both safety and efficacy data. The timing of this interim analysis is expected to be 3 months post the final subject final visit of the AURORA 1 study (i.e., when the last subject reaches Visit 16 of the AURORA 2 continuation study).

## 13.11 Other Evaluations

Not applicable.

## 14. ETHICAL CONDUCT OF THE STUDY

The study will be conducted according to the principles of the World Medical Association's Declaration of Helsinki [22] and the ICH guidelines for GCP [23]. Aurinia will ensure that the study complies with all local, federal, and country regulatory requirements.

The Investigator must ensure the confidentiality of all subjects participating in the study.

All anonymous data remains the property of Aurinia.

#### 14.1 Informed Consent

The ICF used for the study must comply with the Declaration of Helsinki, federal regulations, and ICH guidelines; and must have been approved by the Institutional Review Board (IRB)/Ethics Committee (EC)/Independent Ethics Committee (IEC) prior to use. The Investigator or an authorized associate must explain the nature of the study and the treatment in such a manner that the subject is aware of potential benefits and risks. Subjects must also be informed that participation is voluntary and that they may withdraw from the study at any time, without prejudice. Subjects must be provided sufficient time to consider participation, including discussion with family members prior to signing the ICF. Documentation of the discussion and the date of informed consent must be recorded in the source documentation. After signing the ICF, subjects will be enrolled into the study and assigned the same subject identification number from the AURORA 1 study, that will be used on all subject documentation.

The informed consent can be signed on the Month 12 visit (Week 52/ End of Treatment Visit in the AURORA 1 study).

#### 14.2 Institutional Review Board or EC/IEC

The protocol, any protocol amendments and consent form for the proposed clinical study and any other documents required by the local IRB/EC/IEC must be submitted by the Investigator for review and approval to the IRB/EC/IEC. The Investigator must also ensure that the IRB/EC/IEC reviews the progress of the study on a regular basis and, if necessary, renews its approval of the study per local requirements.

## 15. QUALITY CONTROL AND QUALITY ASSURANCE

The Investigator must ensure that all study-related site source data, study-related documents, and reports will be available, and that the provision of direct access for monitoring and auditing by Aurinia or its designees will be permitted. In addition, the Investigator must ensure that all study-related site source data, study-related documents, and reports will be made available for inspection by the appropriate Regulatory Authority and review by the IRB/EC/IEC.

The Investigator is responsible for notifying Aurinia in advance of an impending regulatory inspection. He/she may request that Aurinia provide support for preparation, if necessary. The Investigator is required to provide updates to Aurinia on the ongoing activities during the inspection, respond to any citations/objectionable findings (i.e., U.S. Food and Drug Administration Form 483) and to share any follow up responses from the Regulatory Authority.

Accurate and reliable data collection will be assured by verification and cross-check of the eCRFs against the Investigator's records by the Study Monitor (source document verification). The Monitor will also review the Investigator's drug accountability records to ensure that the drug supplies are stored and dispensed appropriately. A comprehensive validation program will verify the data and queries will be generated for resolution by the Investigator. Throughout the study, Aurinia or its designates may review data as deemed necessary.

## 16. ADMINISTRATIVE PROCEDURES

## 16.1 Sponsor's Responsibilities

## **16.1.1 Study Supplies**

Sites will be provided with all supplies required to manage this study. This will include but not be limited to the following:

- Investigator file(s) (for filing of all study related documentation).
- Kits for collection, storage, and transportation of applicable samples required for central laboratories. This will also include all applicable guidelines and contact details.
- Contact list of all relevant study personnel.
- eCRF and completion guidelines (or equivalent EDC system).
- Study reference manual.
- All study forms (e.g., SAE, pregnancy, drug accountability, etc.).

#### 16.1.2 Insurance

Aurinia confirms that it carries liability insurance which protects nonemployee physicians or Investigators/study staff against claims for which they may become liable as a result of damages caused by Aurinia- products used in clinical studies. Insurance coverage is not extended to damages that the Investigators or third parties may suffer by reason of acts of commission or omission on the part of such Investigators or third parties and that are not in accordance with accepted common medical practices (*lege artis* procedures). Aurinia will reimburse the subject for all study-related injuries provided that the injury does not arise from the subject's misuse of the study treatment or failure to follow the Investigator's instructions.

## 16.1.3 Study Monitoring

The study will be monitored by representatives of Aurinia (or designee, which may include a contract research organization). If not monitored by Aurinia, documentation of delegation will be described in the Clinical Trial Agreement. It is understood that the responsible Monitor will contact and visit the Investigator regularly and will be allowed, on request, to inspect the various records of the study (eCRFs and other pertinent data) provided that subject confidentiality is maintained in accordance with local requirements.

It will be the Monitor's responsibility to inspect the eCRFs at regular intervals throughout the study (frequency outlined in a separate procedural document), to verify the adherence to the

protocol and the completeness, consistency, and accuracy of the data being entered on them. The Monitor must have access to laboratory test reports and other subject records needed to verify the entries on the eCRF. The Investigator (or his/her deputy) agrees to co-operate with the Monitor to ensure that any problems detected in the course of these monitoring visits are resolved.

## 16.2 Investigator's Responsibilities

## 16.2.1 Reporting and Recording of Data

All required study data must be entered in the eCRF created for the study. Training on the system will be provided to all sites, including instructions on how to address missing data, corrections, query procedures, and electronic signatures. Only individuals who are identified on the authorized signature page may enter/correct data in the eCRF. For those subjects who withdraw before completion of the study, all available efficacy and safety data must be entered in the eCRF. Incomplete or inconsistent data on the eCRF will result in data queries addressed to the Investigator for resolution.

## **16.2.2 Investigator Training**

All Investigators and their study personnel will receive training regarding the study procedures, study treatments, and GCP/regulations specific to the conduct of clinical studies. This training will take place prior to enrollment of the first subject at the study site, and must be documented and filed in the Investigator's Study Site File.

#### 16.2.3 Source Documentation

The Investigator must maintain adequate and accurate records to enable the conduct of the study to be fully documented and the study data to be subsequently verified.

Subject clinical source documents would include subject hospital/clinic records, physician's and nurse's notes, appointment book, original laboratory reports, ECG, X-ray, pathology and special assessment reports, signed ICFs, consultant letters, and subject enrollment logs. These are to be separate and distinct from eCRFs. All data for the study must be available in source documentation, including oral and written communication with the subject regarding the study treatment (including the risks and benefits of the study). The date of informed consent must be recorded in the source documentation.

The Investigator must arrange for the retention of all study documentation (such as eCRFs, research files, and master files) for the duration specified in their respective site contract. The Investigator must keep these documents on file after completion or discontinuation of the study according to local governing guidelines. Archived data may be held electronically, provided that a back-up copy exists and that a hard copy can be generated if required.

| The Investigator must inform Aurinia immediately if any documents are lost, to be transferred to a different facility, or to be transferred to a different owner. | |
|---|---|
| AAAD OD A G (AAAD AAGG 2016 02) AND O | ~ ~ |

# 17. PROCEDURE FOR MODIFICATION OF PROTOCOL OR PREMATURE TERMINATION OF THE STUDY

## 17.1 Protocol Waivers, Deviations and Violations

Protocol waivers shall not be permitted.

The Investigator should not implement any deviation from, or changes of the protocol without written agreement from Aurinia and prior documented approval/favorable opinion from the IRB/IEC of an amendment, except where necessary to eliminate an immediate hazard(s) to study subjects, or when change(s) involves only logistical or administrative aspects of the study. If the Investigator must implement a deviation from, or a change of, the protocol to eliminate an immediate hazard(s) to study subjects without prior written approval, the implemented deviation or change and the reasons for it should be submitted in a timely manner to Aurinia and to the IRB/IEC as required by applicable local requirements.

The Investigator, or person designated by the Investigator, will document and record the preventative and/or corrective measures for any deviation from the approved protocol.

Accidental deviations from the protocol including violations of inclusion/exclusion criteria will be assessed as minor or major on a case-by-case basis. The criteria describing the deviation(s) and how they will be handled will be documented in the SAP.

Any amendment to the protocol requires written approval/favorable opinion by the IRB/IEC prior to its implementation, unless there are overriding safety reasons.

In some instances, an amendment may require a change to the ICF. The Investigator must receive an IRB/IEC approval/favorable opinion concerning the reviewed document prior to administering to study subjects.

## 17.2 Study Termination

Aurinia reserves the right to terminate the study in its entirety or at a site at any time. Reasons for termination may include, but are not limited to, the following: unsatisfactory subject enrollment with respect to quality and/or quantity, site is unable to comply with the requirements of the protocol or GCP, or data recording is inaccurate and/or incomplete.

In terminating the study, Aurinia and the Investigator will assure that adequate consideration is given to the protection of the subjects. Both parties will arrange the procedures on an individual basis after review and consultation and in accordance with the study contract.

## 18. POLICY FOR PUBLICATION AND PRESENTATION OF DATA

Aurinia is committed to the timely communication of data from clinical research trials, following the Pharmaceutical Research and Manufacturers of America principles [24]. Where possible, authorship will be agreed at the beginning of the study. The authors will form a publication committee and this committee will propose and develop appropriate scientific manuscripts or abstracts from the study data. Investigators may not present or publish partial or complete study results individually. Any manuscript or abstract proposed by the Investigators must be reviewed and approved in writing by Aurinia before submission for publication. Names of all Investigators participating in the study will be included in the publication.

The publication committee for a study will comprise of authors selected in adherence with the International Committee of Medical Journal Editors criteria [25] for authorship. If studies are multicenter, it may be appropriate to assign group authorship.

In addition, certain Aurinia employees involved in the design and conception of the protocol, study management and data analysis and interpretation are qualified authors and will be included in the publication committee.

## 19. REFERENCES

- 1. Ward MM. Changes in the incidence of end stage renal disease due to lupus nephritis in the United States, 1996-2004. J Rheumatol. 2009 Jan;36(1):63-7.
- 2. Houssiau FA, Vasconcelos C, D'Cruz D, Sebastiani GD, de Ramon Garrido E, Danieli MG, et al. The 10-year follow-up data of the Euro-Lupus Nephritis Trial comparing low-dose and high-dose intravenous cyclophosphamide. Ann Rheum Dis. 2010 Jan;69(1):61-4. Epub 2009 Jan 20.
- 3. Lee YH, Woo J-H, Choi SJ, Ji JD, Song GG. Induction and maintenance therapy for lupus nephritis: a systematic review and meta-analysis. Lupus. 2010 May; 19(6):703-10. Epub 2010 Jan 11.
- 4. Study WX17801. A prospective, randomized, active controlled, parallel group, multicenter trial to assess the efficacy and safety of mycophenolate mofetil (MMF) in inducing response and maintaining remission in subjects with lupus nephritis (LN). Final report. Victoria (BC): Aspreva Pharmaceuticals Corporation; 2008 May 6. Report No.: 1024493.
- 5. Appel GB, Contreras G, Dooley MA, Ginzler EM, Isenberg D, Jayne D, et al; Aspreva Lupus Management Study Group. Mycophenolate mofetil versus cyclophosphamide for induction treatment of lupus nephritis. J Am Soc Nephrol. 2009 May;20(5):1103-12. Epub 2009 Apr 15.
- 6. Remuzzi G, Ruggenenti P, Benigni A. Understanding the nature of renal disease progression. Kidney Int. 1997;51:2-15.
- 7. Hemmelgarn BR, Manns BJ, Lloyd A, James MT, Klarenbach S, Quinn RR, et al; Alberta Kidney Disease Network. Relation between kidney function, proteinuria, and adverse outcomes. JAMA. 2010 Feb 3;303(5):423-9.
- 8. Trivedi S, Zeier M, Reiser J. Role of podocytes in lupus nephritis. Nephrol Dial Transplant. 2009;24:3607-12.
- 9. Mathieson PW. Proteinuria and immunity an overstated relationship? N Engl J Med. 2008 Dec 4;359(23):2492-4.
- 10. Bao H, Liu ZH, Xie HL, Hu WX, Zhang HT, Li LS. Successful treatment of class V+IV lupus nephritis with multitarget therapy. J Am Soc Nephrol. 2008 Oct; 19(10):2001-10. Epub 2008 Jul 2.
- 11. Miyasaka N, Kawai S, Hashimoto H. Efficacy and safety of tacrolimus for lupus nephritis: a placebo-controlled double-blind multicenter study. Mod Rheumatol. 2009;19:606-15.

- 12. Cortés-Hernández J, Torres-Salido MT, Medrano AS, Tarrés MV, Ordi-Ros J. Longterm outcomes-mycophenolate mofetil treatment for lupus nephritis with addition of tacrolimus for resistant cases. Nephrol Dial Transplant. 2010; 25:393948. Epub- 2010 Jun 10.
- 13. Szeto C-C, Kwan BC-H, Lai FM-M, Tam L-S, Li EK-M, Chow K-M, et al. Tacrolimus for the treatment of systemic lupus erythematosus with pure class V nephritis. Rheumatology. 2008;47:1678-81.
- 14. Uchino A, Tsukamoto H, Nakashima H, Yoshizawa S, Furugo I, Mitoma H, et al. Tacrolimus is effective for lupus nephritis patients with persistent proteinuria. Clin Exp Rheumatol. 2010 Jan-Feb;28(1):6-12.
- 15. Tanaka H, Oki E, Tsugawa K, Nonaka K, Suzuki K, Ito E. Effective treatment of young subjects with pediatric-onset, long-standing lupus nephritis with tacrolimus given as a single daily dose: an open-label pilot study. Lupus. 2007;16(11):896-900.
- 16. Asamiya Y, Uchida K, Otsubo S, Takei T, Nitta K. Clinical assessment of tacrolimus therapy in lupus nephritis: one-year follow-up study in a single center. Nephron Clin Pract. 2009;113(4):c330-6. Epub 2009 Sep 3.
- 17. Tse KC, Lam MF, Tang SCW, Tang CSO, Chan TM. A pilot study on tacrolimus treatment in membranous or quiescent lupus nephritis with proteinuria resistant to angiotensin inhibition or blockade. Lupus. 2007;16(1):46-51.
- 18. Lanata CM, Mahmood T, Fine DM, Petri M. Combination therapy of mycophenolate mofetil and tacrolimus in lupus nephritis. Lupus. 2010 Jul;19(8):935-40. Epub 2010 Apr 13.
- 19. Lee T, Oh KH, Joo KW, Kim YS, Ahn C, Han JS, et al. Tacrolimus is an alternative therapeutic option for the treatment of refractory lupus nephritis. Lupus. 2010 Jul;19(8):974-80.
- 20. KDOQI Clinical Practice Guidelines for Chronic Kidney Disease: Evaluation, Classification, and Stratification, 2002.
  - http://www2.kidney.org/professionals/KDOQI/guidelines\_ckd/p4\_class\_g1.htm. Accessed 2 September 2014.
- 21. Hochberg Y. A sharper Bonferroni procedure for multiple tests of significance. Biometrika. 1988;74(4):800-2.
- 22. World Medical Association Declaration of Helsinki. Ethical principles for medical research involving human subjects. 64<sup>th</sup> WMA General Assembly, Fortaleza, Brazil. October 2013.

- 23. ICH Harmonised Tripartite Guideline.: Guideline for good clinical practice. E6 (R1) 1996 Jun 10.
- 24. PhRMA principles and guidelines: public disclosure of clinical trial results. Pharmaceutical Research and Manufacturers of America [Internet]. 2009 [cited 2009]. Available from: http://www.phrma.org/principles\_and\_guidelines.
- 25. International Committee of Medical Journal Editors [Internet]. Uniform requirements for manuscripts submitted to biomedical journals: writing and editing for biomedical publication [updated 2010 Apr]. Available from: http://www.icmje.org.

## **Appendix 1 Drug Therapy for the Treatment of Hypertension**

Antihypertensive drug therapy for subjects who develop hypertension while on study treatment may include the following:

- Dihydropyridine calcium channel blockers (e.g., amlodipine, nifedipine)
- Alpha-1-adrenergic blocking agents (e.g., doxazosin)
- Alpha-beta-blockers (e.g., carvedilol, labetalol)
- Thiazide diuretics (e.g., chlorthalidone or hydrochlorothiazide)

Excluded Drugs: While the ARBs and ACE inhibitors may also be effective in CNI -associated hypertension, their dose adjustment or commencement is not permitted in this trial (see Section 7.8.1, Prohibited Medications).

## Recommended First and Second Line Therapies for Treatment of Hypertension

Titrate the following according to the timeframe given in the respective drug label:

<u>First Line</u> - select from one of the following:

- Amlodipine, 5 mg daily to achieve BP <140/90 mmHg; titrate to 10 mg daily if satisfactory results not obtained within 2 weeks
- Nifedipine XL, 30 mg daily; titrate to 60 mg and possibly 90 mg daily within 2 weeks
- 12.5 to 25 mg/day of chlorthalidone or hydrochlorothiazide

<u>Second Line</u> - may add from among the following to the first line therapy if a partial response is obtained:

• Labetalol, 100 mg BID; titrate to 200 mg BID, then 300 mg BID

Note: If the BP remains uncontrolled with the above-referenced maximum doses of first and second-line antihypertensive therapies, reduction of study treatment dose may be considered or it may be decided to discontinue study treatment and utilize antihypertensive therapies to achieve control of BP.

If at any time, in the judgment of the treating physician in consultation with the Medical Monitor, the response to treatment is inadequate, the study treatment may be discontinued.

## **Appendix 2** Measurement of Blood Pressure

- 1. Whenever possible, BP measurements should be undertaken by the same study site personnel at each clinic visit.
- 2. Whenever possible, the BP determinations should be undertaken at approximately the same time of day for each study visit and at the same time in relation to prior study treatment ingestion.
- 3. The measurements should be undertaken prior to blood collection.
- 4. Prior to measuring BP, the study subject should be seated in a quiet room for at least 5 minutes, in a chair with his/her back supported and feet comfortably resting on the floor.
- 5. Due to the likelihood each arm can have a slightly different BP, it is strongly encouraged to use the same arm for all measurements, supported at heart level.
- 6. No restrictive clothing should encircle the arm in which BP measurements are determined.
- 7. An appropriately sized cuff will be required wherein the cuff bladder encircles at least 80% of the upper portion of the arm.
- 8. Three serial BP readings will be undertaken with a minimum of 2 minutes between readings and with the cuff fully deflated between each determination.
- 9. The mean of the second and third of these 3 readings will be used as the study day BP value.
- 10. All measurements, along with the calculated mean value, will be recorded in the source documents. The mean of the second and third readings will be calculated within the EDC as the study day result.

## Appendix 3 International Society of Nephrology and the Renal Pathology Society (ISN/RPS) 2003 Classification of Lupus Nephritis

## Class I Minimal mesangial lupus nephritis

Normal glomeruli by light microscopy, but mesangial immune deposits by immunofluorescence

#### Class II Mesangial proliferative lupus nephritis

Purely mesangial hypercellularity of any degree or mesangial matrix expansion by light microscopy, with mesangial immune deposits

May be a few isolated subephithelial or subendothelial deposits visible by immunofluorescence or electron microscopy, but not by light microscopy

## Class III Focal lupus nephritis<sup>a</sup>

Active or inactive focal, segmental or global endo- or extracapillary glomerulonephritis involving <50% of all glomeruli, typically with focal subendothelial immune deposits, with or without mesangial alterations

Class III (A) Active lesions: focal proliferative lupus nephritis

Class III (A/C) Active and chronic lesions: focal proliferative and sclerosing lupus nephritis

Class III (C) Chronic inactive lesions with glomerular scars: focal sclerosing lupus nephritis

#### Class IV Diffuse lupus nephritis<sup>b</sup>

Active or inactive diffuse, segmental or global endo- or extracapillary glomerulonephritis involving  $\geq$ 50% of all glomeruli, typically with diffuse subendothelial immune deposits, with or without mesangial alterations. This class is divided into diffuse segmental (IV-S) lupus nephritis when  $\geq$ 50% of the involved glomeruli have segmental lesions, and diffuse global (IV-G) lupus nephritis when  $\geq$ 50% of the involved glomeruli have global lesions. Segmental is defined as a glomerular lesion that involves less than half of the glomerular tuft. This class includes cases with diffuse wire loop deposits but with little or no glomerular proliferation.

Class IV-S (A) Active lesions: diffuse segmental proliferative lupus nephritis

Class IV-G (A) Active lesions: diffuse global proliferative lupus nephritis

Class IV-S (A/C) Active and chronic lesions: diffuse segmental proliferative and sclerosing lupus nephritis

Class IV-G (A/C) Active and chronic lesions: diffuse global proliferative and sclerosing lupus

nephritis

Class IV-S (C) Chronic inactive lesions with scars: diffuse segmental sclerosing lupus

nephritis

Class IV-G (C) Chronic inactive lesions with scars: diffuse global sclerosing lupus nephritis

## Class V Membranous lupus nephritis

Global or segmental subephithelial immune deposits or their morphologic sequelae by light microscopy and by immunofluorescence or electron microscopy, with or without mesangial alterations

Class V lupus nephritis may occur in combination with class II or IV in which case both will be diagnosed

Class V lupus nephritis show advanced sclerosis

## Class VI Advanced sclerosis lupus nephritis

≥90% of glomeruli globally sclerosed without residual activity

- 1. Weening JJ, D'Agati VD, Schwartz MM, Seshan SV, Alpers CE, Appel GB, et al. The classification of glomerulonephritis in systemic lupus erythematosus revisited. Kidney Int. 2004;65:521-30.
- 2. Weening JJ, D'Agati VD, Schwartz MM, Seshan SV, Alpers CE, Appel GB, et al. The classification of glomerulonephritis in systemic lupus erythematosus revisited. J Am Soc Nephrol. 2004;15:241-50.

<sup>&</sup>lt;sup>a</sup> Indicate the proportion of glomeruli with active and with sclerotic lesions.

<sup>&</sup>lt;sup>b</sup> Indicate the proportion of glomeruli with fibrinoid necrosis and/or cellular crescents.

Indicate and grade (mild, moderate, severe) tubular atrophy, interstitial inflammation and fibrosis, severity of arteriosclerosis or other vascular lesions.

Appendix 4 1997 Update of the 1982 American College of Rheumatology Revised Criteria for the Classification of Systemic Lupus Erythematosus

| Four or More of: | | Definition |
|---|---|---|
| Cri | Criterion | |
| 1. | Malar rash | Fixed erythema, flat or raised, over the malar eminences, tending to spare the nasolabial folds |
| 2. | Discoid rash | Erythematous raised patches with adherent keratotic scaling and follicular plugging; atrophic scarring may occur in older lesions |
| 3. | Photosensitivity | Skin rash as a result of unusual reaction to sunlight, by patient history or physician observation |
| 4. | Oral ulcers | Oral or nasopharyngeal ulceration, usually painless, observed by physician |
| 5. | Arthritis | Nonerosive arthritis involving 2 or more peripheral joints, characterized by tenderness, swelling, or effusion |
| 6. | Serositis | <ul> <li>a) Pleuritisconvincing history of pleuritic pain or rubbing heard by a physician or evidence of pleural effusion</li> <li>OR</li> <li>b) Pericarditisdocumented by ECG or rub or evidence of pericardial effusion</li> </ul> |
| 7. | Renal disorder | <ul> <li>a) Persistent proteinuria greater than 0.5 grams per day (or 0.5 mg/mg by UPCR) or greater than 3+ if quantitation not performed</li> <li>OR</li> <li>b) Cellular castsmay be red cell, hemoglobin, granular, tubular, or mixed</li> </ul> |
| 8. | Neurologic<br>disorder | <ul> <li>a) Seizuresin the absence of offending drugs or known metabolic derangements; e.g., uremia, ketoacidosis, or electrolyte imbalance OR</li> <li>b) Psychosisin the absence of offending drugs or known metabolic derangements, e.g., uremia, ketoacidosis, or electrolyte imbalance</li> </ul> |

| Four or More of:<br>Criterion | Definition |
|---|---|
| 9. Hematologic disorder | a) Hemolytic anemiawith reticulocytosis OR b) Leukopenialess than 4,000/mm³ total on 2 or more occasions OR |
| | c) Lyphopenialess than 1,500/mm³ on 2 or more occasions OR |
| | d) Thrombocytopenialess than 100,000/mm <sup>3</sup> in the absence of offending drugs |
| 10. Immunologic disorder | a) Anti-dsDNA: antibody to native dsDNA in abnormal titer OR |
| | b) Anti-Sm: presence of antibody to Sm nuclear antigen OR |
| | c) Positive finding of antiphospholipid antibodies based on 1) an abnormal serum level of IgG or IgM anticardiolipin antibodies, 2) a positive test result for lupus anticoagulant using a standard method, or 3) a false-positive serologic test for syphilis known to be positive for at least 6 months and confirmed by <i>Treponema</i> |
| | pallidum immobilization or fluorescent treponemal antibody absorption test |
| 11. Antinuclear antibody | An abnormal titer of antinuclear antibody by immunofluorescence or an equivalent assay at any point in time and in the absence of drugs known to be associated with "drug-induced lupus" syndrome |

Abbreviation: ECG = Electrocardiogram.

Sources: Hochberg MC, MD, MPH for the Diagnostic and Therapeutic Criteria Committee of the American College of Rheumatology. Tan EM, Cohen AS, Fries JF, Masi AT, McShane DJ, Rothfield NF, Schaller JG, Talal N, Winchester RJ. The 1982 revised criteria for the classification of systemic lupus erythematosus. Arthritis Rheum. 1982;25:1271-7.

Hochberg MC. Updating the American College of Rheumatology revised criteria for the classification of systemic lupus erythematosus [letter]. Arthritis Rheum 1997;40:1725.

Appendix 5 Systemic Lupus Erythematosus Disease Activity Measure (SELENA-SLEDAI)

| Descriptor | Definition | Points |
|---|---|---|
| Seizure | Recent onset. Exclude metabolic, infectious or drug causes. | 8 |
| Psychosis | Altered ability to function in normal activity due to severe disturbance in the perception of reality. Include hallucinations, incoherence, marked loose associations, impoverished thought content, marked illogical thinking, bizarre, disorganized or catatonic behavior. Exclude uremia and drug causes. | 8 |
| Organic brain syndrome | Altered mental function with impaired orientation, memory or other intellectual function with rapid onset and fluctuating clinical features. Include clouding of consciousness with reduced capacity to focus and inability to sustain attention to environment plus at least 2 of the following: perceptual disturbance, incoherent speech, insomnia or daytime drowsiness, or increased or decreased psychomotor activity. Exclude metabolic, infectious or drug causes. | 8 |
| Visual disturbance | Retinal changes of SLE. Include cytoid bodies, retinal hemorrhages, serous exudate or hemorrhages in the choroid, or optic neuritis. Exclude hypertension, infectious or drug causes. | 8 |
| Cranial nerve<br>disorder | New onset of sensory or motor neuropathy involving cranial nerves. | 8 |
| Lupus headache | Severe persistent headache; may be migrainous but must<br>be nonresponsive to narcotic analgesia. | 8 |
| Cerebrovascular accident | New onset of cerebrovascular accident(s). Exclude arteriosclerosis. | 8 |
| Vasculitis | Ulceration, gangrene, tender finger nodules, periungual infarction, splinter hemorrhages, or biopsy or angiogram proof of vasculitis. | 8 |

| Descriptor | Definition | |
|---|---|---|
| Arthritis | More than 2 joints with pain and signs of inflammation (i.e., tenderness, swelling, or effusion). | 4 |
| Myositis | Proximal muscle aching or weakness associated with elevated creatine phosphokinase or aldolase, or electromyogram changes, or a biopsy showing myositis. | 4 |
| Urinary casts | Heme-granular or RBC casts. | 4 |
| Hematuria | >5 red blood cells per high powered field. Exclude stone, infection or other causes. | 4 |
| Proteinuria | >0.5 g per 24 hours or 0.5 mg/mg UPCR by FMV. New onset or recent increase of more than 0.5 g per 24 hours. | 4 |
| Pyuria | >5 white blood cells per high power field. Exclude infection. | 4 |
| New rash | New onset or recurrence of inflammatory type rash. | 2 |
| Alopecia | New onset or recurrence of abnormal patchy or diffuse loss of hair. | 2 |
| Mucosal ulcers | New onset or recurrence of oral or nasal ulcerations. | 2 |
| Pleurisy | Pleuritic chest pain with pleural rub or effusion or pleural thickening. | 2 |
| Pericarditis | Pericardial pain with at least 1 one of the following: rub, effusion or ECG confirmation. | 2 |
| Low complement | Decrease in CH50, C3 or C4 below the lower limit of normal for testing laboratory. | 2 |
| Increased DNA binding | >25% binding by Farr assay or above normal range for testing laboratory. | 2 |
| Fever | >38°C. Exclude infectious cause. | 1 |
| Thrombocytopenia | <100,000 platelets per mm <sup>3</sup> . | 1 |
| Leukopenia | <3,000 white blood cells per mm <sup>3</sup> . Exclude drug causes. | 1 |

Abbreviations: ECG = Electrocardiogram; RBC = Red blood cells; SLE = Systemic lupus erythematosus.

Source: Bombardier C, Gladman DD, Urowitz MB, Caron D, Chang DH, and the Committee on Prognosis Studies in SLE. Derivation of the SLEDAI: a disease activity index for lupus subjects. Arthritis Rheum. 1992;35:S630-40.

## **Appendix 6** Expanded List of Allowed Concomitant Medications

- Prophylactic therapy for steroid-induced bone loss (calcium with Vitamin D and/or a bisphosphonate).
- Low dose aspirin is allowed for cardiovascular prophylaxis.
- Minor GI AEs (such as nausea, vomiting and diarrhea) may be treated symptomatically (e.g., with loperamide for diarrhea or standard anti-emetics such as metoclopramide or domperidone for nausea and vomiting). Proton pump inhibitors or ranitidine are permitted for dyspepsia or gastric protection. Magnesium or aluminum containing antacids may be used, but should not be taken at the same time as study treatment; such antacids, if required, should be taken either 1 hour before or 2 hours after study treatment.
- Amphotericin or oral nystatin are permitted as infective prophylaxis against fungal infections, and low-dose sulfamethoxazole/trimethoprim is permitted as prophylaxis against *Pneumocystis carinii pneumonia*.
- Granulocyte colony stimulating factor is allowed to manage neutropenia in the presence of major infection (i.e., infections requiring IV antibiotics).
- Oral or IV iron preparations for iron deficiency and/or anemia.
- Erythropoietin is permitted for treatment of severe anemia (hemoglobin <10 mg/dL).
- Cytomegalovirus prophylaxis is permitted for example with oral valganciclovir.
- Acute intermittent administration of NSAIDs for not greater than 7 consecutive days is permitted.
- Lipid-lowering therapies (e.g., statins) will be used as clinically indicated.
- Antimalarials should be prescribed when clinically indicated.
- Angiotensin-converting enzyme inhibitors, ARBs, and aliskerin and other therapies are recommended, as per standard guidelines but if used their dose must be stable throughout the study. In addition subjects must be on a stable dose of ACE inhibitors or ARBs for 4 weeks prior to enrollment.
- In the case of uncontrolled hypertension (systolic BP >165 mmHg or diastolic >105 mmHg on 2 successive measurements), the addition of a diuretic or calcium channel blocker only are permitted, together with dose decreases or

| interruption Pressure. | of | study | treatment | per | the | instructions | in | Section | 7.9, | Increased | Bloc |
|---|---|---|---|---|---|---|---|---|---|---|---|

## **Appendix 7** Summary of Treatment and Food Restrictions

| Treatment | <b>During Treatment</b> | Reason |
|---|---|---|
| Immunosuppressants other than those allowed by protocol | Prohibited | Interferes with study efficacy endpoints |
| Aminoglycosides Amphotericin B Melphalan Ketoconazole | Prohibited | May potentiate toxicity |
| Rifampin | | |
| NSAIDs chronic dosing (>7 consecutive days) | Prohibited | May potentiate nephrotoxicity |
| P-gp substrates | To be monitored | Drug-drug interaction |
| P-gp inhibitors | To be discussed with Medical Monitor | Drug-drug interaction |
| Androgenic steroids Cimetidine Fluconazole, itraconazole Macrolide antibiotics (azithromycin, clarithromycin, erythromycin) Metoclopramide Barbiturates and derivatives Carbamazepine Octreotide acetate Phenytoin Sulfadimidine (intravenous) Theophylline | To be discussed with Medical Monitor | Drugs interfering with Orelvo metabolism |
| ACE inhibitors and ARBs | Change or commencement prohibited | Interfere with primary endpoint assessment |
| Foods Grapefruit and grapefruit juice | Prohibited | May affect the metabolism of Orelvo |

Abbreviations: ACE = Angiotensin converting enzyme; ARB = Angiotensin receptor blocker; NSAID = Non-steroidal anti-inflammatory drug; Pgp- = P-glycoprotein.

















